Study Number: 114-2014-GES-0035

Protocol: 7.0



Study Title: Development of a MR Scanner Capable of Being

Sited in a Neonatal Intensive Care Unit Study Number: 114-2014-GES-0035 Revision/Amendment 7.0

Version Date 25/Sep/2015

### **Confidentiality Statement**

This protocol is provided for conducting a research study. The information contained in this document is confidential and, except to the extent necessary to obtain informed consent or EC/IRB approval, cannot be disclosed unless required by governmental regulation. Persons to whom any portion of the contents of this document is disclosed must be informed that the information is confidential and may not further be disclosed by them.

 DOC1547483 (Rev. 7.0)

Version Date: 25/Sep/2015

Study Number: 114-2014-GES-0035

Protocol: 7.0



Development of a MR Scanner Capable of Being Sited in a Neonatal Intensive Care Unit

> GEHC Study Number: 114-2014-GES-0035 Revision/Amendment: 7.0 Version Date: 25/Sep/2015

# Investigator's Signature Page

Ihereby agree to:

Site Address

- (i) Conduct the investigation in accordance with the agreement, the investigational plan, applicable MHRA or applicable government regulations, and conditions of approval imposed by the reviewing Ethics Committee, IRB or governing regulatory body;
- (ii) Supervise all testing of the device involving human subjects; and

(iii) Ensure that the requirements for obtaining informed consent are met.

| Investigator Signature | Date |
|------------------------|------|
| Print Name | |
| Site Name | |


**Study Number:** 114-2014-GES-0035

Protocol: 7.0



# **Table of Contents**

This document contains the following sections:

| To | pic | | Page |
|---|---|---|---|
| In | vesti | gator's Signature Page | 2 |
| | | of Contents | |
| | | ent and Version Control | |
| | | riations and Terms | |
| | | Synopsis | |
| O | 1.1. | Preliminary Investigations and Justification | |
| | 1.2. | Literature Review | |
| | 1.3. | Pre-Clinical (animal) Trials and Previous Clinical (human) Experience | |
| | 1.4. | Device Risk Analysis | |
| 2. | Res | earch Device and/or Product | 12 |
| | 2.1. | Identification and Description of Research Device/Product | 12 |
| | 2.2. | Regulatory Status | |
| | 2.3. | Risk Category and Rationale | 17 |
| | 2.4. | Device Classification and Rationale | |
| | 2.5. | Device Issuance and Replacement | |
| _ | 2.6. | Disposition of the Device/Product | |
| 3. | • | ectives of Research Study | |
| | 3.1. | Hypothesis | |
| | 3.2. | Justification | |
| | 3.3. | Study Objectives | |
| 4 | 3.4. | Study Endpoints | |
| 4. | | ign of Research Study | |
| | 4.1.<br>4.2. | Type of Research Study Controls and Minimization of Bias | |
| _ | | | |
| 5. | 5.1. | ly Subjects<br>Number of Subjects | |
| | 5.1. | Subject Population | |
| | 5.3. | Protection of Vulnerable Subjects | |
| | 5.4. | Inclusion Criteria | |
| | 5.5. | Exclusion Criteria | |
| | 5.6. | Screening Subjects for Enrolment | |
| | 5.7. | Duration of Enrolment | |
| 6. | Prod | cedures for Research Study | 27. |
| | 6.1. | General Procedures | 27 |
| | 6.2. | Phase 1 (Feasibility) and Phase 2 (Data Collection) | 28 |
| | 6.3. | Per-Subject Procedures | |
| | 6.4. | Unexpected Findings | |
| | 6.5 | Withdrawal and Discontinuation Criteria | 41 |

Protocol: 7.0



| 6.6. | Study Flowchart | |
|---|---|---|
| 7. Trai | ning Plan | 44 |
| 7.1. | Training Plan for Research Device/Product | |
| 7.2. | Training Plan for Protocol | |
| 8. Data | Analysis and Statistics | <u></u> 45 |
| 8.1. | Statistical Analysis Methods | 45 |
| 8.2. | Interim Analysis | |
| 8.3. | Handling of Missing Data | |
| 8.4. | Pass/Fail Criteria of the Study | |
| 9. Othe | er Interim Activities (Qualitative Interim Summaries) | 47 |
| 9.1. | Phase 1 Qualitative Investigator Summary | 47 |
| 9.2. | Phase 1 and Phase 2 End-of-Phase Interim Reports | |
| 10. | Deviations | 47 |
| 10.1. | Management of Protocol Deviations | 47 |
| 11. | Complaint Handling and Adverse Event Reporting | <u>4</u> 8 |
| 11.1. | Foreseeable Adverse Events and Device Effects | 48 |
| 11.2. | Adverse Event Definitions | 49 |
| 11.3. | Management of Adverse Event Reporting | |
| 11.4. | Management of Serious Adverse Event and Unanticipated Adverse | |
| | Effect Reporting | |
| 11.5. | Management of Device Complaints | |
| 12. | Early Termination or Suspension | 51 |
| 12.1. | Criteria for Early Termination or Suspension | |
| 12.2. | Withdrawal of EC Approval | |
| 13. | Ethics Committee (EC) and Regulatory Filings | |
| 13.1. | Regulatory Authority Approval Requirements (Global) | |
| 13.2. | Ethics Committee Approval Requirements | |
| 13.3. | Management of Protocol Revisions/Amendments | |
| 13.4. | Informed Consent and Privacy Requirements | |
| 14. | Data and Quality Management | |
| 14.1. | $\boldsymbol{\varepsilon}$ | |
| 14.2. | Subject De-identification | |
| 14.3. | Subject Pseudonymisation | |
| 14.4. | Completion of Case Report Forms (CRFs) | |
| 14.5. | Record Retention at the Site | |
| 15. | Monitoring Plan | |
| 15.1. | Brief Description | |
| 15.2. | Reference to Approved Monitoring Plan | |
| 16. | Publication Policy | <u>5</u> 5 |
| 17. | ADDITIONAL COUNTRYPECIFIC REGULATORY | |
| REC | QUIREMENTS | 55 |
| | erences | |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Appendix A—Example of Investigator Summary Document | 58 |
|------------------------------------------------------------|------|
| Appendix B-Example of MR Procedure document | 59 |
| Appendix C-Example of Investigational SingleUse Disposable | |
| Swaddle Log | 61 |
| Appendix D-Example of Possible Software Components | 62 |
| Appendix E-Example of MR Scan Log | 64 |
| Appendix F-Example 3.0TNeonatal MRI Investigational Device | User |
| Experience Questionnaire | 65 |
| Appendix G-Example of SingleUse Disposable Swaddle User | |
| Experience Questionnaire | 67 |
| Appendix H: Amendment to Protocol Version 1.0 | 69 |
| Appendix I: Amendment to Protocol Version 2.0 | 70 |
| Appendix J: Amendment to Protocol Version 3.0 | 76 |
| Appendix K: Amendment to Protool Version 4.0 | 80 |
| Appendix L: Amendment to Protocol Version 5.0 | 84 |
| Appendix M: Amendment to Protocol Version 6.0 | 89 |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



## **Document and Version Control**

This section records all changes made to the protocol for a specific study. In the table below, record each and every relevant change by indicating what changes were made.

| Revision | Date<br>(DD/Mmm/YYY/) | Revision Author | Comments/Changes |
|---|---|---|---|
| 1.0 | 28/Oct/2014 | Angela Johnson | Clinical Writer- Initial draft. |
| 2.0 | 03/Dec/2014 | Angela Johnson | Updated name of medical monitor, as detailed in<br>Appendix H: Amendment to Protocol Version 1.0 |
| 3.0 | 04/Mar/2015 | Angela Johnson | Revised to clarify that the primary endpoint of the study is in accordance with Section 2.1 of Annex X of the EU Medical Devices Directive, which species that verificatio of performance and safety across the study cohort is an essential requirement of the study; details local site feed and sleep procedures; and clarifies the duration of the study at planned for 24 months as detailed in Appendix I: Amendment to Protocol Version 2.0 |
| 4.0 | 26/Apr/2015 | Angela Johnson | Revised to clarify per MHRA questions, as detailed in Appendix J: Amendment to Protocol Version 3.0 |
| 5.0 | 15/May/2015 | Angela Johnson | Revised to clarify per MHRA questions, as detailed in Appendix K: Amendment to Protocol Version 4.0 |
| 6.0 | 13/Aug/2015 | Angela Johnson<br>Yvonne Celestial<br>Lisa Augustine | Revised to clarifymodifications made in prior versionas detailed in Appendix L: Amendment to Protocol Version 5.0. |
| 7.0 | 25/Sep/2015 | Angela Johnson | Revised to clarify modifications made in prior version, a detailed in Appendix L: Amendmento Protocol Version 6.0. |

Study Number: 114-2014-GES-0035

Protocol: 7.0



## ABBREVIATION TERMS

CHF Clinical History File CRF Case Report Form

DMP Data Management Plan

EU European Union

FDA US Food and Drug Administration

ICF Informed Consent Form

ISO International Organization for Standardization

MHRA Medicines and Healthcare Products Regulatory Agency

MR Magnetic resonance

MRI Magnetic resonance imaging
NICU Neonatal Intensive Care Unit

PDU Power distribution unit

PNS Peripheral nerve stimulation

RF Radiofrequency

SAR Specific Absorption Rate
SNR Signal to noise ratio
SPR System problem report
SUS System Usability Scale
Tip Training in Partnership

TVA Tip Virtual Assist (Remote Connectivity)

UK Unites Kingdom
US United States

UXS User Experience Scale


**Study Number**: 114-2014-GES-0035

Device/Product GEHC Modality  $\operatorname{MR}$ 

Protocol: 7.0



| STUDY SYNOPSIS | |
|---|---|
| Study Title: Development of a MR Scanner Capable of Being Sited in a Neonatal Intensive Care Unit Study Number. 114-2014-GES-0035 | |
| Research Type Clinical (human) | |
| Brief Description of Study Purpose | |
| This study investigates a novel magnetic resonance imaging (MS) tem designed by GEHfor imaging viable neonate and infantpopulations. This MR system has a smaller size and designatures that may make it more feasible to locate the system in close proximity trare areas for neonates (birth-1 month) and infants (>1 month to two years), such addinical neonatal intensive care units (NICUs) other infant and neonatal care departments | |
| Thisis a two-phase prospective clinical studyevalua investigational MRI device for neonates and infan | |
| • <u>Phase 1</u> - Initial feasibility assessment and optimization study (Phase 1) which may include hardware and software modifications. These studies are guided by a series of MR scanning procedures defined in sequential Sponsor-provided <i>MR Procedure Documents</i> | |
| • <u>Phase 2</u> - Controlled image and data collection study based on Phase 1 results, in which optimized scan procedure(s) according to <i>MR Procedure Document(s)</i> ll be provided at the start of Phase 2 scanning and a fixed hardware and integrated software configuration will be applied for all subjects. | |
| Investigator feedback on scanning conducted under each MR Procedure Documential be documented. Because the device is intended for use in viable neonate and infant populations, clinical data are required that cannot be conducted in any other populations or simulated on non-human models. Clinical images and associated data as well as assessments of image quality, workflow, and usability will be collected. | |
| Images, associated image data, and subject data collected in both phases of this study may be used for future engineering development and activities that support MR product development, including Sponsor-authorized scientific and marketing activities. Summary evaluation of safety and performance from Phase 1 and Phase 2 may be used in support of regulatory submission, including filings for European CE mark. | |
| SponsorName: GE Healthcare (GEHC) Sponsorcontact Yvonne Celestial, Clinical Affairs Project Manager | Address: 283 rue de la Miniere Buc, 78533, FR Telephonæ +33 130709133 E-mail: Marie Yvonne. Celestia l@ge.com |
| Investigator Name(s) Prof. Paul Griffiths, MB, ChB, PhD Academic Unit of Radiology University of Sheffield Floor C, Royal Hallamshire Hospital | Address Glossop Road Sheffield, UK S10 2JF Telephone +44 (0) 114 271 2587 E-mail: p.griffiths@sheffield.ac.uk |

 DOC1547483 (Rev. 7.0) Version Date: 25/Sep/2015

Study Number: 114-2014-GES-0035

Protocol: 7.0



**Device/Product Description:** Small-footprint 3.0T Neonatal MRI investigational device capable of being located in a NICU and its components, including a single-use disposable swaddle, sizing ring, and transport devices. The device design is based on commercially available Optima MR430s 1.5T, Discovery MR750 3.0T, and SIGNA HDx MR technologies and commercial Sponsor-provided patient monitor (Invivo Corp) and site-owned protective devices (e.g. hearing protection and, if necessary, padding or blankets) will be used. **Regulatory Status:** Pre-Market  $\boxtimes$ 3.0T Neonatal MRI investigational device, its components, and its accessories (Single-use disposable swaddle, Sizing ring, and Transport devices) Post-Market **Duration**: The study plans to enrol patients for approximately 24 months. 3200 N Grandview Blvd Address: Research Manager Name Lisa Augustine Warren, Waukesha, WI 53188-1678 Research Project Manager, Global MR Research **Telephone** +1-440-250-9488 E-mail: Lisa.Augustine@med.ge.com Address: 3200 N Grandview Blvd Waukesha, WI 53188-1678 Medical Monitor Name: Jeff Hersh, MD **Telephone** +1-262-366-7295

E-mail:

Jeff.Hersh@ge.com


Study Number: 114-2014-GES-0035

Protocol: 7.0



# 1.1. Preliminary Investigations and Justification

## 1.2. Literature Review

Demand for postnatal magnetic resonance imaging (MRI) examinations in clinical settings is growing rapidly, in part due to recent improvements in neonatal survival rates and antenatal diagnostic imaging. The US Food and Drug Administration (FDA) defines infants (>1 month to 2 years) and neonates (birth to 1 month) by approximate age and weight. <sup>1</sup> In particular, neonatal MRI has become standard clinical care for neurological and orthopaedic applications at many clinical facilities. <sup>2,3,4,5</sup> Despite this increasing application of MRI to very young subjects, MRI has not been specifically optimized for imaging infants and neonates outside of a few limited research settings. <sup>6</sup> The challenges of neonatal MRI imaging have been extensively documented, <sup>5,4,6,7</sup> leaving significant room for improvement in MRI scanning of neonates to make MRI more practical and comfortable for these vulnerable subjects and their care providers.

MRI is useful for examining neurological disease in the developing brain of young subjects, and MRI also serves a key diagnostic role for a variety of other conditions and abnormalities in developing neonate and infant anatomy. The clinical manifestations of neurological disease are more subtle during early neurological scanning in infants and neonates, and many neural structures that are central to the adult human brain cognitive function are functionally silent in the infant. <sup>8</sup> This poses unique challenges for applying MRI effectively in this population. MRI systems have also been used for orthopaedic, thoracic, and abdominal exams in the first hours of life with good results, though there remains significant room for improvement and optimization of these systems for neonates and infants. <sup>9</sup> In a variety of anatomical regions, high-quality images have been attained with good spatial resolution, signal-to-noise ratio, and tissue contrast using standard clinical MRI protocols in infant and neonate subjects housed in the NICU environment, but the logistics of transport and safety for these subjects remains challenging in most clinical facilities. <sup>9</sup>

In preterm neonates, there is an even more pronounced disconnect between adult and neonatal MR image characteristics, resulting in significant risks associated with misinterpreting MR images resulting from using scanning techniques optimized for adult or older paediatric subjects. <sup>8</sup> Advances in antenatal diagnosis of brain, spine, and body abnormalities as well as diagnostic imaging for specialized conditions, such as ischemic encephalopathy, that rely on MR imaging systems have increased demand for postnatal MRI. <sup>10,8,11</sup> Thus, there is a growing need for high-resolution MR images of the neonatal and infant brain, along with numerous possible clinical and research applications of such imaging.

For neonatal MRI, the vast majority of clinical care facilities use a conventional commercial whole-body MRI system with standard, commercially available coils, though custom-built systems and systems that integrate commercially available incubators have been documented. <sup>12,13,14</sup> Because of the advantage of neonatal MRI, a growing number of clinical facilities are considering installing dedicated neonatal imaging systems that are optimized both logistically, in terms of location relative to the NICU and other infant/neonatal care departments, and in terms of subject care. <sup>15</sup> Recently, a small profile 1.5T MR system has been built by Cincinnati Children's Hospital Medical Center for neonatal MRI and is sited in the neonatal intensive care unit at that institution. <sup>13</sup>

In contemporary clinical practice, there is a growing unmet need for MRI imaging systems that are specifically designed for use in neonatal and infant populations. Though off-label use

Study Number: 114-2014-GES-0035

Protocol: 7.0



of MRI systems approved for adults does occurs in some clinical settings, MRI is still not accessible to the majority of neonates and infants in the current paradigm, and the current trend is away from off-label use of adult devices on infants and neonates. <sup>2</sup> Furthermore, the hardware and software developed for adults is being applied to neonates, often in a suboptimal manner that could involve yet unknown risks and reduce performance in this vulnerable population. <sup>2</sup> There are also notable risks involved in transporting infants from a neonatal intensive care unit (NICU) to a radiology department for MRI, both logistically and medically. <sup>16</sup>

The development and regulatory approval of dedicated MRI systems for neonates and infants may make MRI more widely available to these populations in clinical care settings. The potential advantages of dedicated neonatal MRI systems may include overall reduced cost and site demands, lower acoustic noise, improved ease of access, and reduced medical risk to the neonate. <sup>16</sup> This study investigates a dedicated MRI system developed by the Sponsor for imaging viable neonate and infant subjects.

# 1.3. Pre-Clinical (animal) Trials and Previous Clinical (human) Experience

Research and clinical use of MR imaging has been widely documented in scientific literature over the past three decades, including research as early as the 1980s. <sup>17,18,19,20</sup>
Recommendations have also been made by the American Academy of Neurology and Child Neurology Society <sup>10</sup> to help guide clinical practice when imaging preterm and term infants, stating that "MRI holds great promise; however, this imaging modality and others that may be soon developed must become more infant friendly, and imaging strategies should be developed to provide maximum information in minimum time." Extensive scientific literature exists to support the safety and effectiveness of MRI executed by properly trained operators for neonate and infant populations; <sup>21,22,23,24</sup> however, the physiologic differences in the neonate and infant brain compared to adults leaves room for optimization of MR hardware and software to produce improved results in these populations. <sup>25</sup>

GEHC has not previously conducted clinical studies using the 3.0T Neonatal MRI investigational device under study. A second study using this device in the United States (US) is currently being planned.

# 1.4. Device Risk Analysis

#### 1.4.1. Risks

The 3.0T Neonatal MRI investigational device is intended for use in neonates and infants, and its components and accessories used in this study are based on similar commercial systems labelled for use in patients aged greater than 2 years of age and manufactured by the Sponsor, and these devices have undergone non-clinical qualification and risk assessments conducted by the Sponsor. Participating in this study involves some risks that are unique to the design of the scanner and population (neonates and infants), as described Section 11.1 Foreseeable Adverse Events. This section lists possible foreseeable adverse events and device effects, but actual occurrences of these risks are uncommon and are not anticipated to occur frequently, if at all, in this study. While serious adverse events can occur in MRI exams in rare cases, typically with adverse events occurring as a result of failure to correctly follow routine site MR safety procedures for scanning, no serious adverse events are anticipated in this study.

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



Subjects participating in research MRI scanning in this study are not expected to be at increased discomfort or risk beyond that posed by other standard of care MRI devices. The investigational single-use disposable swaddle is a medical device that is expected to have risk comparable or less than routine MR padding, blanketing, and/or other transportation devices. During the study, the subject will be transported and cables or other devices may be disconnected or connected, which could cause discomfort or interruption of care. The investigator is responsible for ensuring minimal disruption of normal care during the study.

### 1.4.2. Benefits

Subjects are not expected to directly benefit from participating in this study, and no diagnostic or other care will be determined based on research MR scanning in this study.

### 2. RESEARCH DEVICE AND PRODUCT

## 2.1. Identification and Description of Research Device/Product

## 2.1.1. 3.0T Neonatal MR Investigational Device

The investigational device being studied is a 3.0T Neonatal MRI device intended for use in neonates and infants. The device has a small size profile that makes it capable of being sited in a NICU or other neonatal and infant care units. This device includes an MR system and its hardware and software components is a whole body magnetic resonance scanner designed to support high resolution, high signal-to-noise ratio and short scan times. It is indicated for use as a diagnostic imaging device to produce axial, sagittal, coronal, and oblique images and proton spectra of the body of neonates and infants. It is specifically designed so that the system is able to be sited in or near NICUs, including having smaller overall dimensions and weight compared to conventional commercial whole-body MRI scanners. This reduces the structural and space requirements for housing the device. Many components of the device are based on engineering designs used in the commercially released Optima MR430s 1.5T, the Discovery MR750 3.0T, and the SIGNA HDx Family of MR systems.

The device is also designed with accessories to make transport of the neonatal subject from the bedside to the MR scanner more efficient. Image data produced by the 3.0T Neonatal MRI investigational device is capable of reflecting the spatial distribution or molecular environment of nuclei exhibiting magnetic resonance. Due to the nature of this research study, the device will not be used diagnostically for the purpose of this study, and study scans are conducted for research purposes only.

# 2.1.2. 3.0T Neonatal MRInvestigational Device Components and Initial Configuration

The configuration of the device at the beginning of the study includes the central hardware and software components, as follows:

## System Hardware Components

1. **3.0T Magnet**: The device uses a 3.0T magnet based on GEHC's commercially released Optima MR430s 1.5T musculoskeletal MR system. The device's 3.0T magnet, unlike predecessor 1.5T magnets, is designed to increase image signal-to-noise ratio which is important in imaging this subject population in order to maximize tissue contrast in the images.

Study Number: 114-2014-GES-0035

Protocol: 7.0



- 2. **17.86cm (diameter) Bore:** The bore is the opening in the center of the device in which the subject is placed during MR scanning. Color-coded landmarking controls are used to assist in positioning subject anatomy in the bore.
- 3. Gradient Coils and Gradient Drivers (70 mT/m gradient strength and 300 T/m/s slew rate: The gradient system used in the device is based on the combined technologies of the Optima MR430s 1.5T and SIGNA HDx series MR systems with adapted HDx gradient driver technology. Magnetic gradients are slight changes in the main magnetic field due to three electrically controlled orthogonal coils oriented in the x, y, and z directions of the scanner. These gradients are involved in signal localization and imaging plane selection (axial, sagittal, coronal, and oblique).
- 4. Radiofrequency (RF) System he RF transmitter consists of an exciter (synthesizer), power amplifier, and transmitting/receiving coil. The exciter design is based on the commercially released Discovery MR750 3.0T system, and the amplifier is a new design specifically made for this device. The RF device consists of a coil, pre-amplifier, and signal processing system. The transmitting and receiving coil is a single channel sixteen rung "birdcage" coil (inner surface accessible to the subject). The RF transmits proton-exciting energy into tissues, and subsequent proton relaxation energy emission is detected by receiver RF coils. This data is processed into MR images. The closer fit to specific neonate anatomy is intended to improve RF signal detection in order to improve image quality.

**Transport Cart (Table)** The small profile transport cart docks to the MR scanner table for bedside-to-MR transport within space-limited care areas for neonates and infants, such as NICU environments.

### **System Software Components**

All of the pulse sequences, post-processing, and visualization software are based on, and are similar in design and function to other commercially released software for GEHC MR scanners. Software components that may be variably used in this study are detailed in <a href="Appendix D - Example of Possible Software Components">Appendix D - Example of Possible Software Components</a>. These include the following primary software components:

- 1. Pulse Sequences Pulse sequences are software sets of RF (and/or gradient) magnetic field pulses and time spacing's between these pulses that can be used in conjunction with magnetic field gradients and MR signal reception to produce MR images. These software sets are installed on the system and are thereafter available for use with specific operator-set parameters. The pulse sequences being studied are similar in design and function to commercially available pulse sequences. The type of pulse sequence and parameter settings that dictate the timing and shape of the pulses provide the operator control over the image contrast. In most clinical MR exams, images are acquired with multiple pulse sequences with various settings, allowing clinicians to compare and distinguish tissues and abnormalities. The site may also provide phantoms for study use.
- 2. MR PostProcessingand Visualization Software: Post-processing and visualization software are software modules and/or algorithms that manipulate the images for purposes such as, but not limited to, changing the characteristics of the images and generating parametric maps and related reports.

Study Number: 114-2014-GES-0035

Protocol: 7.0



Additionally, services and accessories that are intended to work with the device may be used in this study, as follows:

### **System Accessories**

- 1. **Straps**: The straps secure the patient to the table during the scan.
- 2. **Sizing guide (sizing ring tool)** The sizing ring tool is a horseshoe-shaped component used to ensure the patient (with all required accessories) will fit into the bore of the MR device.
- 3. **Neonate MR Padding**Special padding for neonates and infants has been designed to work with the investigational device.
- 4. **System Sevice Tools/Phantoms (Simulations)** Phantom images are simulations of human scanning that can be completed without a real human subject in the magnet bore. During the study, the Sponsor and the investigator may generate and run phantom imaging procedures on the device. Phantoms may be provided for training, education, engineering, and optimization purposes.
- 5. **Remote Connectivity.** The device is capable of remote connectivity through the Training in Partnership (TiP) Virtual Assist (TVA) program, which offers secure data connections between a Sponsor representative and the device user for use in training, trouble-shooting, and real-time image quality optimization during scanning.

## 2.1.3. Single-use Disposable Swaddle

The single-use disposable swaddle is an investigational medical device that is a soft, pliable, blanket-type accessory with Velcro® closures intended for swaddling infant or neonate subjects on both sides and feet before, during, and immediately after MR scanning. The swaddle has been designed for patient transfer and positioning and allows the infant to be securely positioned and immobilized during the lift and transfer process. The swaddle also provides line management for any gating wires and/or tubes that may be attached to the infant and to any devices. The swaddle is disposable and intended for single-use only. It is considered to be an accessory to the MRI system that contains the following key components:

- 1. **Velcro® closures** Internal and external closures secure the infant/neonate using Velcro® straps.
- 2. **Textile material**: Swaddles are constructed of soft, dual-layer, pliable, blanket-type textile materials.
- 3. **Backboard**: The backboard is a non-disposable component that can be optionally used with the single-use disposable swaddle to stabilize larger subjects.

Protocol: 7.0





Figure 1 – Image of swaddled neonate entering the 3.0T Neonatal MRI investigational device bore (top left) and views of soft, duallayer textile swaddleshowing Velcr® closures

# 2.1.4. Other MREquipment

The Sponsor may also provide other commercial MR equipment required to conduct the study, including:

- a. physiologic motion synchronization devices,
- b. protective padding,
- c. hand-held metal detector,
- d. patient monitoring equipment (i.e. Invivo Corp monitor), and
- e. other commercial MR accessories

There may be other commercial equipment provided to the investigational site(s) as part of this study. All commercial equipment provided to the investigational site will be documented in the Sponsor's Clinical History File (CHF) in the *Device Accountability Log*nd communicated in writing to the investigational site. The intent to use any other commercial MR accessory devices that are not explicated described in the protocol procedures during clinical scanning procedures will be documented in the Sponsor-provided *MR Procedure Document* do records will be retained in the *Device Accountability Log* 

Study Number: 114-2014-GES-0035

Protocol: 7.0



## ExpressionPatient Monitor (Invivo, Corp; Orlando, FL, US)A

Expression Monitor (Invivo Corp.) – This is an MR Conditional patient monitor system labelled for use in neonate and infant populations that can remain in the magnet room during scanning. Depending on workflow, this can also be sited near the operator console for patient monitoring during the MR scan.

Invivo Corp patient monitor will be used during study procedures to monitor subject vital signs, body temperature (on the Expression Monitor using a single-use sensor in the MRI scan room), and  $O_2$  saturation.

## 2.1.5. Device Configuration Management

Throughout Phase 1 (Feasibility and Optimization) part of this study, the configuration of the device, including hardware and software components, may be altered for engineering research and optimization purposes to gai*m vivo*human data about the optimal device configuration. For Phase 2, single device configuration will be used.

The Sponsor will ensure that changes in device configuration will:

- a. Not increase risk classification of the study;
- b. Not increase subject and/or operator risk;
- c. Be released internally by the Sponsor prior to release to the investigational site;
- d. Be communicated in writing to the Principal Investigator (PI) and stored in the Sponsor's Clinical History File (CHF); AND
- e. Be accompanied by appropriate training materialselated to changes in device configuration, if determined to be necessary by the Sponsor or upon request of the PI.

**Note**: No changes in device configuration will be implemented that are not communicated in writing by the Sponsor to the Principal Investigator and stored in the Sponsor's Clinical History File (CHF) as part of the evice Accountability Lognd maintained in the Site Regulatory Binder

For changes in device configuration, the Principal Investigator assumes responsibility for:

- a. Providing confirmation of device configuration changes and ensuring that these are stored in the Site Regulatory Binder
- b. Ensuring that Sonsor-provided communications or electronic copies thereof are stored in the Site Regulatory Binder
- c. Ensuring that Study Staff are trained and documentation is retained of such training for Sponsorprovided training materials and, as necessary, changes device configuration and records.

**Note**: The PI may request additional training from the Sponsor if necessary, at his or her discretion. All training will be documented. In addition to Spons**pr**ovided training, the PI and designated study staff may perform phantom scanning not using human subjects for the purpose of training and retraining staff members at any time during the study.

# 2.2. Regulatory Status

The 3.0T Neonatal MRhvestigational devices a pre-market magnetic resonance diagnostic device and its accessories and omponents are not yet cleared for commercial use (pre

Study Number: 114-2014-GES-0035

Protocol: 7.0



market). In the United Kingdom (UK), the use of the device is subject to regulation by the Medicines and Healthcare Products Regulatory Agency (MHRA), in compliance with the Medical Devices Regulations of 2002 (transposition of European Medical Device Directive 93/42/EEC concerning medical devices, including Articles 3, 15, Annexes VIII and X).

The Expression MRI patient monitoring system (Invivo, Corp; Orlando, FL, USA) provided by the Sponsor for use in this have received CE mark for commercial use and are labelled for use in neonate and infant populations. All patient monitoring equipment will be used in accordance with its labelled indications, including meeting all conditions for MR scanning for MR Conditional devices.

## 2.3. Risk Categoryand Rationale

The MRI device used in this study uses static magnetic field strengths <4.0T, which are widely accepted to pose minimal risks to typical adults, children, and infants/neonates, as detailed in the US FDA Guidanc@riteria for Significant Risk Investigations of Magnetic Resonance Diagnostic Device\*\*and contemporary medical literature\*\*<sup>26,27</sup> During this study, subjects will encounter routine risks of transport outside of their regular care environment, which are considered mitigated to levels as low as reasonatphyacticable (ALARP) by design of the device and attendance of medical personnel throughout the subject's transport and study procedures. The 3.0T Neonatal MRhvestigational device under study uses a 30T static magnetic field The Sponsor'&iskManagement procedures demonstrate that risks have been appropriately mitigated according to ISO 14971, icompliance with regulatory requirements set forth by the Medicines and Healthcare Products Regulatory Agency (MHRA), in compliance with the European Medical Device Ditieve 93/42/EEC.

### 2.3.1. MR Safe, Conditional, and Unsafe

Some medical devices placed into surgically or naturally formed cavities of the human body (implants) or other device or objects outside of the body may be allowed into the MR environment, however, MR lexaminations may be contraindicated in patients with some types of passive or active implants at cannot be safely allowed in the MR environment the these procedurs and the site MR safety policy are followed, the risks associated with devices and objects within the MRI environment are considered to be no greater than routine clinical MRI scanning.

ASTM F25035tandard Practice for Marking Medical Devices and Other Items for Safety in the Magnetic Resonance Environmentovides terminology for classifying Inether implants pose

Study Number: 114-2014-GES-0035

Protocol: 7.0



potential hazards to patients in the MR environment that is recognized in the European Union and United States Food and Drug Administration (FDA), [1],[2] as follows:

| Label | Description (typical use) |
|----------|---------------------------|
| MR | |
| or<br>MR | MR Safe |
| MR | MR Conditional |
| MR | MR Unsafe |

**Note:** If the level of MR compatibility of the device in question is not known (not presented on the device label) or the device identity is not able to be determined, then an implantable ice should be considered MR Unsafe for the purposes of this study, with the exception of dental devices/fillings, surgical clips, and surgical staples determined to be safe for MRI scanning by a physician investigator.

Special care should be taken iMRI with metal objects typically found on neonates and infants, such as umbilical cord clips and identification bands. The local site MR safety policy should be followed when determining if these devices are safe for MRI.

### 2.4. Device Classification and Rationale

In the United Kingdom (UK), the investigational 3.0T Neonatal MRI investigational device and its components and accessories used in this study are considered a Class IIa medical device per the European Medical Device Directive Annex IX, Rule 10. The Single-use Disposable Swaddle and its components and accessories are considered to be a Class I medical device per the European Medical Device Directive Annex IX, Rule 10.

In the UK, the Expression MRI patient monitoring systems (Invivo, Corp; Orlando, FL, USA) are considered Class IIa medical device per the European Medical Device Directive Annex IX, Rule 10.

# 2.5. Device Issuance and Replacement

#### 2.5.1. Issuance and Installation

The Sponsor will ship to the study site and install the investigational 3.0T Neonatal MRI investigational device. The Sponsor will provide single-use disposable swaddles and

<sup>[1]</sup> Establishing Safety and Compatibility of Passive Implants in the Magnetic Resonance (MR) Environment. US Food and Drug Administration (FDA). August 21, 2008, updated April 6 2011.

<sup>&</sup>lt;sup>[2]</sup> European Union (EU) Directive 2004/40/EC and 2008/46/EC

Study Number: 114-2014-GES-0035

Protocol: 7.0



necessary hardware and software components and accessories for the investigational system.

If not already owned by the investigational site, the Sponsor may provide each site with Sponsor-owned Expression (Invivo Corp) patient monitoring systems labelled for use in neonate and infant populations according to MR Conditional labelling. Unique identifying information will be recorded for both Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and a copy of this information will be stored in the Sponsor-provided and site-owned devices used in this study and s

### 2.5.2. Medicinal and Biologic Product Administration and Delay

No clinically indicated medical care will be additionally administered or delayed for any subject due to study participation. No medicinal agents (including sedatives), biologically active agents, or contrast agents not required for the subject's clinical care outside of this study will be administered for the purpose of this study, with the exception of routine sweet solutions ('sweeties') which may be used during the study period if prescribed by a physician.

Subjects that received sedatives or other clinically indicated medicinal or contrast agents as part of their regular clinical care may be included if there are no extensions of administration or delays to administration of clinically indicated medications (including treatments required to end sedation) as a result of study participation. Sedation may not be extended for the purpose of this study.

#### 2.5.3. Future and Concurrent Use of Devices

This study is being conducted for engineering development and regulatory submission (including CE mark in the EU) of an investigational medical device and its components and accessories. After the device is CE marked, the device and/or its components may be used concurrently in other research activities in the EU under EC/IRB approved protocols, subject to, and required to adhere to, applicable local laws and regulations, and to the requirements of the Sponsor for device accountability. Any concurrent research activity will also be required to receive approval from the Sponsor and the institutional EC/IRB at the investigational site(s). This information may also be used for regulatory purposes in other countries outside of the EU. If the device is used in other countries, future and concurrent use will adhere to applicable laws and regulations.

## 2.5.4. Research Device Labelling

The device and related components will be labelled as an investigational device in accordance with local regulatory requirements in the UK. Labeling for investigational device(s) shall be provided by the Sponsor in a format approved by the Sponsor and consistent with local regulatory requirements at the investigational site.

### 2.5.5. Maintenance and Replacement

During this study, the Sponsor will be conducting engineering optimization and ensuring that the device(s) operate as intended, which may involve maintenance or replacement of hardware or software components of the device(s) and device accessories at the investigational site(s). To this end, Sponsor-authorized personnel may:

Study Number: 114-2014-GES-0035

Protocol: 7.0



- a. Access device(s) in-person or remotely (such as through TVA/TiP or other secure remote connection) for quality control, trouble-shooting, training, real-time image optimization, to collect system configuration and system log files, or other purposes required for device maintenance, installation, de-installation, and/or system data collection;
- b. Conduct phantoms (simulated non-human) scans;
- c. Repair or replace the device or any of its components;

The Principal Investigator (PI) assumes responsibility for promptly reporting any device-related adverse events or product complaints observed by the PI or study staff to the Sponsors Clinical Affairs Project Manager (CAPM).

## 2.5.6. Security for Investigational Devices

- 1. **Single-use DisposableSwaddles:** Single-use disposable swaddles and non-disposable backboards will be uniquely and sequentially numbered and stored in a locked cabinet accessible to study staff. The investigational site will log the use and disposal of each swaddle (Appendix B). Swaddles are intended for use with the investigational device under this protocol, and swaddles may not be used outside of a Sponsor- and EC/IRB-approved study protocol. Each swaddle may be used only once, and may only be used on a single subject.
- 2. **Power Distribution Unit**: The Sponsor may lock the Power Distribution Unit (PDU) to secure the investigational device if changes are made to the device configuration requiring additional study staff training or maintenance.
- 3. **Host Computer**. The host computer will accessible to authorized study staff, including the PI and trained scan operators, with a Sponsor-provided username and password.
- 4. **Security for the MR Environment** The investigational device will be housed in a secured environment that meets the Sponsor's engineering specifications for device installation. This area and the entrance to the scan room will accessible only to the PI and trained study staff. The Principal Investigator assumes responsibility for meeting all investigational site and Sponsor requirements for securing the device.

# 2.6. Disposition of the Device/Product

When scanning under EC/IRB approved study protocols, the following actions will be conducted:

- a. The Sponsor will ensure that the device(s) and its components are dispositioned according to the contractual agreement reached between the investigational site and the Sponsor, in accordance with applicable local laws and regulations.
- b. The Investigator will ensure that used disposable components, such as used swaddles, will be handled according to the investigational site(s) standard procedures for disposal of biomedical waste.
- c. The Investigator will ensure that unused disposables and other non-disposable equipment provide by the Sponsor (including any Sponsor-provided Invivo Corp Expression patient monitor, hand-held metal detectors provided by the Sponsor, and the non-disposable backboard for the swaddles) are returned to the Sponsor.

Study Number: 114-2014-GES-0035

Protocol: 7.0



### 3. OBJECTIVES OF RESEARSTUDY

## 3.1. Hypothesis

There is no statistical hypothesis being tested in this study. Descriptive statistics will be used to provide summary evaluations of performance and safety data.

## 3.2. Justification

This study is being done in two parts to optimize and collect data from a new MRI device for use in neonates and infants, the 3.0T Neonatal MRI investigational device. The first part of this study is being conducted to demonstrate the feasibility and safety of attaining diagnostic quality images and data using the 3.0T Neonatal MRI investigational device in neonates and infants with various hardware and software configurations. The second part of this study is being conducted to collect images and associated data in neonates and infants from a fixed hardware and software configuration of the 3.0T Neonatal MRI investigational device in support of regulatory activities in the European Union (EU), including CE mark. MR system log files containing operating parameters relative to safety and performance calculations will be systematically collected throughout the study for all subjects. Summary performance and safety evaluations from both parts of the study may be disclosed to regulatory agencies as part of this study.

## 3.3. Study Objectives

## 3.3.1. Primary Objective(s)

To evaluate the safety and performance of the device by collection of images and associated data using the 3.0T Neonatal MRI investigational device that demonstrates the feasibility of use in clinical neonate and infant populations.

## 3.3.2. Secondary Objective(s)

To collect per-subject image quality, usability, workflow, and transport data.

To collect usability information for each device configuration (pMR Procedure Document

To optimize device use and configurations, including ftware and hardware components functionality with MRaccessories and performance factors.

## 3.3.3. Exploratory Objectives:

To record persubject information, including clinical and demographic data.

To collect image data related to clinical follows conducted (if applicable) for engineering and device optimization purposes.

# 3.4. Study Endpoints

### 3.4.1. Primary endpoints

For bothPhase 1 and Phase 2, primary endpoints will be recorded as:

• Collection of MR images and associated data per quotas (Section 5.1.1 - Quotas by Anatomic Region)

Study Number: 114-2014-GES-0035

Protocol: 7.0



- Performance will be determined by summary proportions of images determined to be of evaluable or non-evaluable diagnostic quality
- Safety will be determined by summary rates of adverse events

## 3.4.2. Secondary endpoints

- MR image quality evaluation(s), per-phase as follows:
  - o Phase 1 and 2 all subjects): Overall image quital rated on a 15 Likert scale
  - Phase 1 Qualitative evaluation and optimization (Summary Report) provided by PI, as per applicable MR Procedure Document
  - o Phase 2-Evaluations as described in the Procedure Document
- Persubject Transport and swaddlingimes and data
- Persubjectworkflow and transportinformation
- Persubjectformative and summative usability information (<u>Appendix F-Example</u> 3.0TNeonatal MR Investigational DeviceUser Experience Questionnair <u>Appendix G-Example</u> of SingleUse DisposableSwaddle System User Experience Questionnaire
  - Phase 1-Collected as onsite Sponsor study staffobservations
     (may be completed by Sponsor staff trained on the stpdytocoland/or onsitestudy staff)
  - Phase 2-Collected by onsite assessments by thecan operator (must be completed by trained site study staff)
- Number and type(as determined by Sponsor engineeringpresentativebased on investigator device complaint reports) f device issues, as follows:
  - Technical Issues (causeby operator error)
  - Malfunctions (device did not perform as intended)

## 3.4.3. Exploratory endpoints

- Perpatient medical conditions, information, and demographics as described in the procedure sections
- Phase 1only—Engineering/optimization images and associated image data from clinically indicated MRI followup for unexpected findings

### 4. DESIGN OF RESEARCHUBY

# 4.1. Type of Research Study

## 4.1.1. Study Type

This is atwo-phase, single-site, open-label, prospective research tudy involving human neonate and infant subjects This study is designed as a twphase clinical trialwith a feasibility and optimization phase (Phase 1) and controlled image collection study (Phase 2)

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



Phase 1 is being conducted to optimize and calibrate the device for subsequent data collection in Phase 2 of this study. Both parts may be used for regulatory submission purposes, including CE mark and submissions to other global regulatory authorities in other countries.

| Open-Label<br>Blinded | | All MR scarconfigurationsare known to researchers andubjects |
|---|---|---|
| Double-Blinded | | |
| Singlesite<br>Multi-site | $\boxtimes$ | There is one investigational site |
| Randomization<br>Procedure | | |
| Not randomized | | Randomization is not required, as theiseno comparative hypothesis testing |
| Single arm<br>Comparator | | There are nocomparison or control group |
| Parallel<br>Crossover | | |
| Prospective | $\bowtie$ | Subjects are enrolled and then undergo study procedures |

# 4.1.2. Rationale for Two-PhaseStudy Design

This study is being conducted in two phases, as follows:

Phase 1: The first phase (Phase 1) is a feasibility and optimization assessment that cannot be conducted in any other population and is designed to allow collection of clinical image and associated data as well as to assess image quality, workflow, and usability in human subjects. The results from Phase 1 will be considered in deciding whether to continue to Phase 2 and, if Phase 2 is conducted, the most appropriate device configuration. Phase 1 data is not primarily intended for regulatory submission but may, if determined necessary by the Sponsor, be disclosed to regulatory authorities in support of regulatory submission.

<u>Phase 2</u>: Phase 1 will be followed by a sequential second phase (Phase 2) to collect human images and data intended to as sample images and associated per-subject data for use in regulatory submissions.

Images and data from both Phase 1 and Phase 2 may be used to support future engineering activities.

### 4.2. Controls and Minimization of Bias

The following bias control methods are being employed in this study:

a. <u>Selection bias</u> will be limited by consecutively enrolling subjects meeting the inclusion/exclusion criteria

Study Number: 114-2014-GES-0035

Protocol: 7.0



- b. <u>Spectrum bias</u> will be limited by using a population expected to be representative of the general population at the investigational site, without regard for gender, race, or ethnicity.
- c. Reader bias will be limited by ensuring that evaluators and readers making performance assessments are separate radiologists (not the PI or neonatologist).

### 5. STUDY SUBJECTS

## 5.1. Number of Subjects

Subjects will be enrolled in two phases, to achieve thirty (30) datasets in Phase 1 (Feasibility and Optimization) and up to five (5) datasets in Phase 2 (Data Collection) for a total of thirty-five (35) total evaluable datasets in both phases.

To achieve the target of 35 datasets, a total maximum of 60 subjects may be enrolled per the sample size calculation shown in Section 8.1.1 – Sample Size Determination. The minimum number of patients possible will be used to achieve the target number of evaluable datasets.

## 5.1.1. Quotas by Anatomic Region

The expected 35 evaluable datasets required for this study are set forth in the quota detailed in Table 2 by anatomical region. There is only one anatomical region for this study.

Table 2- Number of evaluable image datasets

| | Approximate number of evaluable datasets required (n) | |
|---|---|---|
| Anatomic Region | Phase 1<br>(Feasibility and<br>Optimization) | Phase 2<br>(Data Collection) |
| Neurological(Head/Neck/Spine) | 30 | 5 |

<sup>\*</sup>n = approximate total number of evaluable datasets

The Sponsor may choose to end either Phase of the Study when adequate datasets are achieved, based on determination made by the SponsAny such determination that would limit enrolment within a phase and/or individual quota group will be communicated in writing to the investigational siteAny such limitations that apply only within a single quota group do not constitute termination of the study.

## 5.1.2. Special Considerations for Enrolment

The following special considerations apply to bject enrolment in both Phase 1 and Phase 2

 Incomplete Datasets: Datasets may be incomplete due to factors such as noise, sequence failure, or patient movemenDatasets determined to be incomplete or non-evaluable by the investigator will not be counted towards the total required datasets for the purposes offetermining quotafulfilment (per protocol population,) but these will be reported in the total patient proliment in the study final report

Study Number: 114-2014-GES-0035

Protocol: 7.0



(intent-to-treat population). Both complete and incomplete images and data will be stored and provided to the Sponsor for engineering purposes.

2. Changes to Quota Requirements during the Study: The Sponsor reserves the right to change quota or Phase dataset number requirements at its discretion and for any reason within the set patient enrolment maximum. The Sponsor will notify the investigational site in writing of any changes in enrolment quotas.

## 5.2. Subject Population

Viable neonate and/or infant subjects that meet the inclusion and do not meet the exclusion criteria will be enrolled.

## 5.3. Protection of Vulnerable Subjects

## 5.3.1. Vulnerable Subjects

This study involves a vulnerable population (viable neonates and infants), per ISO 14155:2011 that defines a vulnerable subject as any individual whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate. This definition includes children, such as the neonates and infants included in this study, which would otherwise require consent from a legally authorized representative acting in their best interests.

This study is being conducted to collect images and data on a device intended for use in neonates and infants that could not be otherwise conducted without using this vulnerable population. The Sponsor has conducted previous internal testing using phantoms to evaluate the safety of the device for use on humans.

Protection of these vulnerable subjects is imperative and the following safeguards will be employed:

- a. Only viable, living neonates and infants will be included in this study;
- b. No neonates of uncertain viability or nonviable neonates will be included in this research;
- c. Individuals engaged in the research will have no part in determining the viability of a neonate, and all such determinations will be made according to the standard clinical practice at the investigational site.

### 5.4. Inclusion Criteria

Subjects will be included that are:

- 1. Currently admitted for treatment or observation at the investigational site at the time of enrolment;
- 2. In the weight range less than  $5.0 \text{ kg} (< 5.0 \text{ kg}^1)$  and more than  $0.5 \text{ kg} (> 0.5 \text{ kg}^2)$ ;
- 3. Viable neonates (birth to 1 month of age) or infants (>1 month to two years of age);<sup>3</sup>
- 4. Able to safely undergo an MRI scan, as determined by medically qualified personnel;

<sup>&</sup>lt;sup>1</sup> <5.0 kg is considered equivalent to <5000.00 g

<sup>&</sup>lt;sup>2</sup>>0.5 kg is considered equivalent to <500.00 g

<sup>&</sup>lt;sup>3</sup> 1 month is considered equivalent to 30 days; 2 year is considered equivalent to 729 days or less

Study Number: 114-2014-GES-0035

Protocol: 7.0



- 5. Have parent(s), guardian(s), or legally authorized representative(s) willing and able to provide written informed consent for the subject's participation;
- 6. Are of appropriate size and shape to fit into the bore of the magnet, inclusive of all monitoring equipment, if any, necessary for the subject's routine clinical care based on standard of care measurement methods, in accordance with site policies:
  - a. Maximum width (shoulder-to-shoulder measurement) less than eighteen (18 cm).
  - b. Maximum length (head-to-foot measurement) less than sixty (60) cm.

## 5.5. Exclusion Giteria

Subjects will be excluded that:

- 1. Have parent(s), guardian(s), or legally authorized representative(s) that require that they accompany the subject into the MR environment that have contraindications to the MR environment or would otherwise be put at undue risk or discomfort, as determined by medically qualified personnel;<sup>4</sup>
- 2. Have any ferrous or electrical items or non-removable medical devices that are not compatible with MR scanning (including devices labelled as MR Unsafe, MR conditional for which the scanning conditions are not met, or without MR safety labelling that does not satisfy site MR safety requirements) that may pose hazards in the MR scanning or MR environment, in the opinion of the Principal Investigator or medically qualified personnel in accordance with the site's MR Safety policy;
- 3. Have any contraindications or could otherwise be expected to experience detrimental effects to safety, well-being, or medical care, as determined by the Principal Investigator or medically qualified personnel in accordance with the site's MR Safety policy;
- 4. Require any scheduled standard of care procedures that are expected to be adversely impacted by participation in this study, in the opinion of the principal investigator or medically qualified personnel; and
- 5. Have been previously enrolled AND undergone any study procedures under the current study protocol (i.e. the same subject cannot undergo study procedures, including swaddling and/or MR scanning, more than once).

# 5.6. Screening Subjects for Enrolment

## 5.6.1. Subject Recruitment

Subjects that are expected to meet the site's MR Safety Policy criteria and any additional supplemental safety policies criteria recommended by the investigator (as per the exclusion criteria) and are otherwise eligible for inclusion will be recruited through a neonatologist, neonatologist fellow, or study staff authorized through written delegation at each investigational site, in accordance with EC/IRB policy.

<sup>&</sup>lt;sup>4</sup> If it is not safe for the parent or guardian that wishes to accompany the subject into the MR environment, the parent or guardian may opt not to accompany the subject. In this case, the subject would not be excluded. Subjects would be excluded if it is determined to be potentially unsafe for a parent or guardian to accompany a subject into the MR scan suite, and the parent or guardian is not willing to allow the subject to be scanned alone while he/she waits in another area of the hospital.

Study Number: 114-2014-GES-0035

Protocol: 7.0



## 5.6.2. Screening for Enrolment

Potential subjects will be identified by the Principal Investigator or other qualified site staff. Informed consent will be obtained for those subjects who agree to participate in the study. Subjects will then be screened for enrolment to ensure the subject is eligible to participate per the inclusion/exclusion criteria, as per the judgement of medically qualified personnel.

Subjects who do not qualify based on inclusion/exclusion criteria will be considered screen failures.

Once a subject is determined to be eligible per the inclusion/exclusion criteria including providing written informed consent, the subject will be considered enrolled and assigned a subject number.

### 5.7. Duration of Enrolment

The study plans to enrol patients for approximately 24 months.

### 6. PROCEDURES FOR RESELASTUDY

#### 6.1. General Procedures

### 6.1.1. Quality Control Scans

The study staff conducting the investigational MR scans (scan operator) will conduct regular Quality Control scans using phantom imaging according to the MR system Operator Manual. The results of Quality Control scans will be stored at a secure location at the investigational site and may be reviewed by the Sponsor.

#### **Phantom Scanning**

The investigator and/or Sponsor representatives may execute phantom scans that simulate human scanning for the purposes of training, troubleshooting, or other engineering optimization purposes at any time during the study.

#### Specific Absorption Rate (SAFS)cans

The device is equipped with a predictive SAR model designed to conservatively limit actual SAR exposure in research subjects. The predictive SAR model used on the system is detailed in the technical documentation for the Neonatal MRI device. Each scan session will include sequences designed to generate a range of actual SAR data, which is stored in system logs and subsequently collected by Sponsor engineering representatives. Throughout the study, system log files containing experimentally generated SAR data will be routinely collected, along with relevant clinical datasuch aspatient weight (as described in subsequent protocol section), necessary forfuture evaluation of the system's predictive SAR model versus actual clinical datain the infant/neonate population.

#### MR ScanSession Log

In order to account forall MR scarsessions using the investigational MR system he scan operator will maintain a daily MRS can Session Logicause this investigational MR scanner may be used for concurrent research protocols, the MR Scan Session Logical E-

Study Number: 114-2014-GES-0035

Protocol: 7.0



<u>Example of MR Scan Log</u>) may also contain entries from other approved studies. For this study, the log will include:

- a. the GEHC-issued study number,
- b. subject number,
- c. date of imaging
- d. MR Procedure Document version number, in applicable
- e. anatomy imaged
- f. comments, if applicable

The log will continue as long as the investigational MR device is housed at the site, and will only be discontinued when all EC/IRB-approved studies are completed and the investigational MR device(s) is/are removed from the investigational site.

**Note**: Allhuman scans for this study, scans done for any otherctive EC/IREapproved studies using this device, and other norclinical scans (i.e. phantom scarfs research, service/maintenance, or training) will be logged. This is done so that the log is consistent with the internal log inside of the system for engineering purposes The log may contain other columns required by other concurrent protocols and some fields may be marked as not applicable (N/A) for other concurrent protocols.

# 6.2. Phase 1 Feasibility) and Phase 2 (Data Collection)

Phase 1 of the study will be conducted to collect feasibility data and optimize the MR system. Throughout the term of the Study, the Sponsor will communicate with the PI and Study Staff as requiredfor device optimization. The Sponsor will provided Procedure Docume sto the site, and the PI or delegate will complete and return qualitative Investigator Summary within approximately 3 businessdays after the procedures described in the current MR procedure document have been completed. The Sponsomay provide additional sequentially numbered MR Procedure Document is significant.) iterative adjustment the procedure for subsequent MR scanning.

Phase 2 will be conducted to collestample images and associated data for regulatory submission. While hardware and software may be modified throughout Phase 1, a fixed hardware and software configuration will be used for all Phase 2 scanning seed on the results of Phase 1 MRP rocedure Document (se) III be provided to the site and used consistently in all Phase 2 scanning

During both phases, remote TVA connectively feature will be available to scan operators for the purposes of training, troubleshooting, and retime image quality optimization during phantom and clinical proceduresTheTVAfeature limits remote connectivity so that no scanning can be initiated without scan operator confirmation.

#### 6.2.1. MR Procedure Documents

At the beginning of the study (prior to initial scanning) the Sponsor will provide an interpretable of the site of

Sponsorprepared MR Procedure Documentail include the following items:

• MR Procedure Document rsion

Study Number: 114-2014-GES-0035

Protocol: 7.0



- Date of Document
- Estimated number of subjects that will be subject to a particular MR Procedure Document.
- Comments/Specific Instructions for procedures to be performed
  - Additional Sponsor-Requested Assessments of performance characteristics on a 1-5 Likert Scale<sup>5</sup>, which may include:
    - Assessments of performance
    - Overall image quality
    - Image contrast
    - Artefacts
    - Fat/water homogeneity
    - Signal-to-noise ratio (SNR)
    - Reconstruction software performance
    - Optimization of application packs (pulse sequence and postprocessing software)
    - Usability
    - And/or other assessments

**Note**. The investigator is responsible for completing only the assessments indicated by the current version of the MR Procedure Document he investigator should ensure that all study staff completing assessments are aware any changes.

- Effective Date that the specified study procedures should begin (i.e. begin on or after this date)
- Name and signature of Sponsor Engineering Representative
- Name and signature of Sponsor Clinical Affairs Project Manager

Each MR Procedur Document will be assigned a unique, consecutive numerical, Version number (e.g. 1.0, 2.0, 3.0, etc.).

No human MR scanning for this Study will be conducted outside of a Sporaeuthorized MR Procedure Documen Phantom scanning may be conducted for training and maintenance purposes without a MR Procedure Document Scanning that is not compliant with MR Procedure Document ill be considered a deviation and ill be reported according to Section 9.1—Management of Protocol Deviations

*Note* For image quality assessme, scores of 3, 4, or 5 will be considered diagnostic quality, and scores of 1 and 2 will be considered non-diagnostic quality.

<sup>&</sup>lt;sup>5</sup> Likert Scale of 45, where:

<sup>1 =</sup> Very Poor

<sup>2 =</sup> Poor

<sup>3 =</sup> Neutral

<sup>4 =</sup> Good

<sup>5 =</sup> Excellent

Study Number: 114-2014-GES-0035

Protocol: 7.0



## 6.2.2. Qualitative Investigator Summary (Phase 1 only

The PI will completen qualitative *Investigator Summar*(<u>Appendix A-Example of Investigator Summar</u>) documents within approximately 3 business days of completion *MR Procedure Document* The Qualitative Investigator Summary will include:

- Consecutively numbered Investigator Summary Number
- Version number of MR Procedure Document ( ing discussed
- Qualitative Comments related to results
- Comments/Suggestions for optimization of future study procedures (i.e., workflow, scanning, usability)
- PI or delegate's name, signature, and date completed

All completed *Investigator Summaries* ill be submitted by the PI or delegate to the Sponsor's *ClinicalAffairs Project Manages* ho will sign and date each document to confirm receipt and store a copy of the document in the Sponsor's Clinical History File (CHF).

# 6.3. Per-Subject Procedures

## 6.3.1. Pre-MR ScanningActivities

## MRPre-Screening

To verify that subjects with necessary medical equipment present can safely fit into the study device bore with normal airflow and without contact, subjects will be verified to be of acceptable size for study MR scanning using the Sponsor-provided sizing tool ('horseshoe" shaped ring) with necessary attached medical equipment prior to removal from the normal clinical care environment.

**Note**: The sizing tool is a study device that may only be used after written informed consent for participation has been attained.

The study staff will then ensure that the subject and any person(s) accompanying him or her into the MR environment satisfy all applicable site MR Safety Screening requirements.

If the subject is determined not be of appropriate size, not to meet MR Safety Screening policies at the site, or is discharged from clinical care at the investigational site prior to MR scanning, the subject will be withdrawn from the study.

## Duration of Active Enrolment (for AE/SAE reporting purposes)

Subjects may be transported to the MR suite before or after removal from their incubator, crib, or other standard of care bedding.

Subjects will be considered actively enrolled (for AE/SAE reporting purposes) in the study on a per-subject basis from the time that the Sponsor-provided horseshoe-shaped sizing tool is used to measure subject size (the first study procedure of MR Pre-Screening). It is mandatory that the sizing ring is used for all subjects before other study procedures to ensure that the subject is of proper size for the MR bore.

Study Number: 114-2014-GES-0035

Protocol: 7.0



Active enrolment will be considered to end on a per-subject basis upon the later of:

- a. The time that the subject is returned to his or her standard of care clinical environment and all Sponsor provided devices are removed from the subject, including Sponsor-provided swaddle, protective padding, and all other study devices.
- b. After active enrolment ends, images and data about any standard of care follow-up or other medical care resulting from unexpected findings may still be accessed observationally and collected by the Sponsor for research purposes.

## Pre-Study Feed and Sleep Procedures

Per the applicable standard of care procedures required at the investigational site, each participating neonate or infant subject will be allowed adequate feed and sleep to ensure minimum disruption of care during MRI scanning, as follows:

- a. The subject will be either breast or bottle fed by or in the presence of the parent/legal guardian.
- b. The subject will be placed in a position that is relaxed and comfortable, with the expectation that it will be reasonably possible for the subject to sleep through the MRI scan.

### Swaddling Subjects and Use of Protective Padding

If used, unique identification number of the Sponsor-provided single-use disposable swaddle will be documented and noted on the swaddle log (Appendix C – Example of Single-Use Disposable Swaddle Log), and the following data will be collected during swaddling:

- Was a Sponsor-provided swaddle used (Y/N). If no, explain why not.
- Was other hospital-provided swaddling (e.g., blankets) used (Y/N); explain why
- Swaddle ID number
- Time of subject placement in the swaddle (on 24 hour clock)
- Swaddled shoulder circumference (in either swaddle or other padding)
- Shoulder-shoulder length before swaddling
- Description of when swaddling occurred (e.g., diapering, bathing, feeding or changing, etc.)
- Was backboard used (Y/N). If yes, explain why used

Subjects should be placed into the Sponsor-provided swaddles by trained study staff according to the instructions provided by the Sponsor. Subjects may be placed in the Sponsor-provided swaddles either immediately before transport to the MR suite or at an earlier time that will minimize subject discomfort, such as during routine feeding, bathing, or diapering. Efforts should be made to place subjects in the Sponsor-provided swaddles as close as possible to the time of MR scanning unless this presents a potential hazard or undue discomfort to subjects. If a swaddle is not used, the subject should be snuggly placed in blankets provided by the investigational site, as such to prevent direct contact between the subject and the walls of the 3.0T Neonatal MRI investigational device (the bore) during scanning.

Study Number: 114-2014-GES-0035

Protocol: 7.0



The site should follow the Sponsor's operator manual for specifications and application of padding to the subject prior to scanning, and padding provided by the Sponsor should be utilized for all subjects. At the discretion of the Principal Investigator or medically qualified delegate, the site may also apply necessary additional site-provide padding along with Sponsor-provided padding.

### General Method for Recording Temperature

Subject body temperature will be recorded at defined intervals before, during, and after scanning as detailed in the following sections. In the MR suite and during scanning, MR Safe Invivo Expression monitors should be used to determine temperature and other vital signs.

## Pre-Transport Subject Information

The following pre-scan session subject information will be recorded for all subjects:

- gender
- age since birth(days for subjects aged ≤30 days and months for subjects aged >30
- gestational age (for subjects ≤30 days old)
- infant or neonate status (neonate = birth to  $\leq$ 30 days; infant  $\geq$ 30 days to  $\leq$ 2 years)
- Pre-transport temperature body temperaturejust before leaving the incubator or crib, measured according to the standard clinical practice at the investigational site as follows:
  - o temperature measurement value
  - o device type (record standard of care device), and
  - o anatomical area of measure (specific area of skin surface)
- head circumference
- weight on day of scan
- Additional Sponsor-Requested Assessments:
  - Blank areas will be included for these assessments (10 blank "Assessment Title" lines with associated 1-5 Likert scales) will be provided on the CRF to accommodate Sponsor-requested elements that may be specified for each MR Procedure Documenthe investigator is responsible for being aware of any additional elements required by each MR Procedure Documents rision number. The investigational site(s) will be notified of any additional instructions for completing comments, and will be responsible for completing the comments field as instructed after appropriate training and instruction has been provided by the Sponsor.
- Investigator comments
  - The investigator is encouraged to make additional comments on any atypical or exceptional conditions of the subjects, including but not limited to pertinent medical history or known deformity.

## Pre-ScanSubject Transport

The subject will be transported to the MR suite either before or after swaddling (whichever is less disruptive to the subject's care, in the opinion of the study staff) from his or her standard clinical care environment. The following parameters will be recorded about subject transfer to the MR scanning location:

 Version Date: 25/Sep/2015

Study Number: 114-2014-GES-0035

Protocol: 7.0



- Transport mode into MR suite (subject moved by incubator/crib to MR suite or subject moved by transport cart/table)
- Time of removal from incubator/crib (on 24 hour clock)
- Number of staff required to transfer (departing incubator/crib; arriving MR)

The transfer table will be docked to the MR scanner and advanced to centre the anatomy of interest (known as 'land-marking') relative to the MR scanner. Transport is considered to end when the table is docked and the subject is advanced into the magnet bore.

#### Pre-scan Environmental Condition

Immediately prior to the first scan series, the following environmental conditions in the MR scanning room will be recorded:

- Scan room temperature
- Number of personnel required to transport the MR table from the MRI preparation room into the scan room, dock the cart/table to the MR scanner and position, landmark, and advance the subject into the magnet bore

#### Protective Devices/Procedures

All subjects require mandatory hearing protection that provides a minimum of 22 dB attenuation prior to MR scanning (ear plugs or a combination of ear plugs and ear muffs, in accordance with site MR Safety Polices).

Use of the horseshoe-shaped sizing ring to verify that subjects can safely fit into the bore of the MR device is mandatory immediately prior to scanning.

The scan operator or delegate will ensure that the subject meets the criteria for MR scanning according to the site MR Safety Policy. In addition, the study staff may screen subjects and accompanying person(s) for presence of ferrous metallic objects using a hand-held metal detector, under the direction of the principal Investigator or delegate. If new information shows that the subject does not meet the site MR Safety Policy requirements, the subject will be withdrawn.

In neonate and infant populations, special care should be taken to check umbilical or limb security devices that may have metal parts that are not safe for MRI scanning. Check if the infant or neonate has any umbilical clips or name bands with metal parts for MR safety before entering the MRI suite; remove them if deemed MR unsafe and it is safe to remove these per the standard clinical practice at the site. Special care should be taken to remove all metal objects from subjects and persons accompanying the subject prior to initiating MR scanning. If objects or devices that are not safe for MRI scanning are not able to be removed safely, the subject should be withdrawn from the study.

Protective padding shall be used on all subjects according to the device's operator manual and it is preferred that the Sponsor-provided protective padding is used. If the site uses site-provided protective padding for a particular subject, the reason for not using the Sponsor-provided protective padding will be documented.

Study Number: 114-2014-GES-0035

Protocol: 7.0



## **Preparation for Scanning**

Immediately before initiating the scan, ensure that the Expression Monitor (Invivo) is connected and monitoring vital signs, including but not limited to body temperature and O<sub>2</sub> saturation. Once acclimated to the scan environment, the following scanning information shall be recorded by the scan operator, including the following:

- Pre-scanning baseline temperature ody temperaturemeasurement made with Invivo Expression Monitor (Invivo) s follows:
  - o the time (minutes) allowed for acclimation once in the magnet bore before taking the temperature measurement
  - o temperature measurement value
  - o anatomical area of measure (specific area of skin surface).

The study staff will set the alarm level on the Expression Monitor (Invivo) to trigger at 0.5°C above the pre-scanning baseline temperature.

## 6.3.2. MR ScanningProcedures

## Monitoring Subjects during MR Scanning

During MRI scanning, subjects will be monitored in real-time using a properly functioning Expression MRI Patient Monitor (Invivo, Corp; Orlando, FL, USA). The subject will be observed all times during the MR scan by a qualified medical professional (nurse, neonatologist, and/or other medical doctor qualified for neonatal/infant care) on the study staff who shall remain in the magnet room with the subject during scanning. The observing staff should remain in a position where they can readily observe the subject and monitor and, if necessary, contact the scan operator during the scanning session.

Aconservative threshold for body temperature alarm is selected, as such that body temperature change is sufficient to trigger an alarm (0.5°C above the pre-scanning baseline temperature) is not in itself considered a clinically significant risk to patients; these patients will be evaluated by a medically qualified member of the study staff for any other possible signs or symptoms and they will determine whether an AE has occurred as per the standard procedures described in Section 11 – Complaint Handling and Adverse Event Reporting.

If a body temperature alarm on the monitor is triggered at any time during scanning, the study staff should stop the scan series. Then, the following elements will be documented as part of study data for each such alarm occurrence:

- o the time of a larm
- o Alarm Temperature the body temperature at time of a larm, based on body temperature measurement made with the Expression Monitor (Invivo), as follows:
  - temperature measurement value
  - anatomical area of measure (specific area of skin surface).
- o the time it takes to return to pre-scanning baseline temperature (minutes/seconds)

**Note.** In the event that thebaby's body temperature does not return to level at or below theorescanning baseline temperature within the studycanning period (not to exceed 60 minutes from first localizer to end of scanning patient scanning will be discontinued (if collected, the patient's data collected up until this time may still be used for study purposes, and pestanning information may still be recorded about the patient)

Study Number: 114-2014-GES-0035

Protocol: 7.0



- any conditions observed that possibly contributed to temperature rise, such as swaddling, environmental conditions, distress, or scanning conditions? (Y/N, if yes explain)
- o decision to continue the scan session (do not continue after first alarm)? (Y/N)
- Continuing Temperature
   the body temperature at the time of scanning was continued using an Expression Monitor (Invivo) s follows:
  - temperature measurement value
  - anatomical area of measure (specific area of skin surface).

Amedically qualified investigator should evaluate each patient to determine if it is safe to continue scanning once the patient's body temperature returns to pre-scanning baseline temperature or lower in the event of an alarm. If an alarm is triggered more than once during a single scan session, scanning will be discontinued. If collected, the patient's data collected up until this time may still be used for study purposes, and post-scanning information may still be recorded about the patient.

## Subject MR Sanning Procedures

The total time starting from the start of the first localizer to the time at the end of the last scan will not exceed sixty (60) minutes. Additional time may be required for setup and removal of the patient.

The scan operator will:

- a. enter the subject's anonymized ID number in the "Subject Name" and "Subject ID" field in the MR scanner's user interface.
- b. enter the subject's weight in the MR scanner's user interface.

In addition to the scan operator, a member of the study staff cleared to enter the MR magnet room will remain in the MR suite at all times when a subject is present in order to assist the scan operator should an emergency situation arise

## MR Scanning Information

For each scanning session, the following scanning information shall be recorded by the scan operator, including the following:

- MR Procedure DocumeNersion Number
- Phase of Scanning (Phase 1 or Phase 2)
- Subject number
- Date of scanning
- Was the subject sedated for standard of care reasons prior to scanning (Y/N)
- Time and type of clinically indicated sedative administration

**Note**: No sedatives will be administered for the purpose of this study. Check yes only if the subject was previously administered clinically indicated sedative(s) within the last 24 hours prior to scanning.

 Start and End time of scanningdetermined bytime just prior to first localizeand time at end of lastscan (on 24 hour clock)

Study Number: 114-2014-GES-0035

Protocol: 7.0



- Scan operator name and signature
- Anatomy scanned (i.e. neurological (head/neck/spine) Was subject fed before (<1 hour) prior to scanning? (Y/N)
- Did subject require pacifying during scan? (Y/N)Were there any repeat scans done due to motion artefacts caused by subject voluntary motion? (Y/N)
- Were there any recoverable system errors or failures during the scanning session?
   (Y/N) If Yes, please describe.
- Comment: Describe any image features which may have negatively affected the image quality including items such as, but not limited to, artefacts, tissue contrast, noise etc.
- Additional Sponsor-Requested Assessments
  - Modifiable CRF fields (10 blank "Assessment Title" lines with associated 1-5 Likert scales) will be provided on the CRF to accommodate Sponsorrequested elements that may be specified for each R Procedure Document
    - The investigator is responsible for being aware of any additional elements required by each *MR Procedure DocumeNe* rsion number.
    - The investigational site(s) will be notified of any additional instructions for completing comments, and will be responsible for completing the comments field as instructed after appropriate training and instruction has been provided by the Sponsor.
- Investigator Comments
  - The investigator is encouraged to make additional comments on any atypical or exceptional events that occur during subject scanning.
  - During the study, the Sponsor may provide additional instructions for recording specific types of conditions or information in the comments field at its discretion as part of an MR Procedure Document
  - The study staff will be responsible for completing the comments field as instructed in the applicable *MR Procedure Docume(nt*) dicated by version number) after appropriate training and instruction has been provided by the Sponsor.

In Phase 1, the Sponsor's engineering representative, if present, may optionally record any applicable comments on a dedicated CRF page.

#### MR Scannerlssues

<u>Issues that occur during the scanning session</u>: In the event of recoverable issues during the scan session:

- a. the scan operator will generate an issue report according to the instructions provided by the Sponsor,
- b. Data may be collected from the MR scanner by the Sponsor's authorized engineering representative.

**Note**: AnySponsorengineer involved at the sitevill betrained on the clinical protoco These Sponsorengineers are qualified to answer technical questions about the device, build not be authorized toprovide training, retraining, or answer study conduct questions raised by
Study Number: 114-2014-GES-0035

Protocol: 7.0



study staff, such as issues with informed consent or other protocol issues/questions. Study conduct questions that are non-technical in nature should be referred to the Clinical Affairs Project Manager. Device use, installation, operation, maintenance, and other technical questions may be addressed with on-site engineers.

<u>Non-recoverable malfunctions</u>: Non-recoverable malfunctions will be considered those that are not resolved by the scan operator rebooting/resetting the system. In the event of a non-recoverable MR system malfunction:

- a. the scan session will be stopped,
- b. the subject will be removed from the MR environment and returned to their standard of care environment,
- c. the equipment will be assessed by the Sponsor, and
- d. The Sponsor must authorize that the device may be used prior to scanning additional clinical subjects.

## 6.3.3. Post-scanning MR Procedures

## Post-scanning Subject Information

Post-scanning information will be recorded for all subjects:

- Postscanning temperature
  Body temperature, immediately before removal from the
  MR scanner (postcan body temperature,)body temperature measurement made
  with an Expression Monitor (Inviva)nd anatomical area of measure (specific area of
  skin surface).
- *Final temperature*Body temperaturemeasuredafter transport andjust before the subject isplaced into the routine careenvironment, as follows:
  - o temperature measurement value
  - o device type (record standard of care device), and
  - o anatomical area of measure (specific area of skin surface)

*Note*. It is preferred that the same method as used for the transport Temperature

- End of Enroment Time: Time when the patient is returned to the clinical careea and all Sponsorprovided device components (i.e., Swaddle, Invivo monitor, pads, etc.) have been removed from the subject.
- AdditionalSponsorRequested Assessments
  - CRF fields (10 blank "Assessment Title" lines with associated likert scales) will be provided on the CRF to accommodate Sponsæquested elements that may be specified for eachMR Procedure Document
    - The investigator is responsible for being aware of any additional elements required by each MR Procedure DocumeNt rision number.
    - The investigational site(s) will be notified of any additional instructions for completing comments, and will be responsible for completing the comments field as instructed after appropriate training and instruction has been provided by the Sponsor.

#### • Comments

o The investigator is encouraged to make additional comments on any atypical or exceptional events that occur during subject scanning. During the study, the Sponsor may provide additional instructions for recording specific types of conditions or information in the comments field at its discretion as part of

Study Number: 114-2014-GES-0035

Protocol: 7.0



an *MR Procedure Document* he study staff will be responsible for completing the comments field as instructed in the applicable *Procedure Document* (indicated byversion number) after appropriate training and instruction has been provided by the Sponsor

#### Post Scan Environmental Conditions

At the end of the last scan series when the scan operator enters the scan room to remove the subject from the MRIevice, the scan operator will record

- Scan room temperature
- Number of personnel required to remove subject from the scanner and undock the cart/table from the MR scanner and transport the MR table out of the scan room and into the MRI preparation room.

#### Post ScanOperator Assessments

For each subject, a designated study staff member present during the MR scan session will complete the usability survey for all applicable device components (Appendix F – Example of 3.0T Neonatal MRI Investigational Device User Experience Questionnaire; Appendix G – Example of Single-Use Disposable Swaddle User Experience Questionnaire). More than one study staff may collaborate to complete these surveys, but only one survey form should be completed based on the consensus between all participating study staff. The Sponsor's representative may also collect observational comments during human scanning.

#### 6.3.4. Evaluations

#### Performance Evaluation

Image sets will be labelled according to subject identification number. Images will be evaluated as evaluable (diagnostic) or non-evaluable (non-diagnostic) by two evaluators, and then evaluable images will be read for image quality by a separate reader, as shown in Figure 2.

**Study Number**: 114-2014-GES-0035

Protocol: 7.0





**Figure 2**– Flowchart of performance evaluation. Determination of evaluable/non-evaluable for diagnostic purposes will be used as the primary performance measure. All secondary Image Quality Assessments will be descriptively summarized.

MR image datasets for each subject will be evaluated twice by two delegated radiologists serving as image evaluators (Evaluator 1 and Evaluator 2) as:

- Evaluable (Diagnostic Quality) 6, or
- Non-evaluable (Non-Diagnostic quality).

The evaluations and printed name and signature of the image evaluator(s) will be recorded to an Evaluator CRF. In the event that the two evaluators (Evaluator 1 and Evaluator 2) disagree on whether an image is evaluable or non-evaluable, a third medically qualified reader (Reader 1) will arbitrate to provide an evaluable/non-evaluable decision, which will be recorded to the Reader CRF and treated as the final decision for the image set.

## Image Quality Assessments

All evaluable images will be further examined by a single reader (Reader 1) that may be the PI or a qualified delegated radiologist for image quality on a 1-5 Likert Scale, 7 as follows:

Overall image quality

*Note* For image qualityassessment, scores of 3, 4, or 5 will be considered diagnostic quality, and scores of 1 and 2 will be considered nondiagnostic quality.

<sup>&</sup>lt;sup>6</sup> An image set may be considered of diagnostic quality if it contains images suitable for diagnosis (not all images views are typically required to be diagnostic based on specific scanning circumstances, so long as applicable views necessary for diagnosis are present)

<sup>&</sup>lt;sup>7</sup> Likert Scale of 1-5, where:

 $<sup>1 = \</sup>text{Very Poor}$ 

<sup>2 =</sup> Poor

<sup>3 =</sup> Neutral

<sup>4 =</sup> Good

<sup>5 =</sup> Excellent

Study Number: 114-2014-GES-0035

Protocol: 7.0



**GE** Healthcare

- Image contrast
- Presence of artefacts
- Signal to noise ratio (SNR)
- Tissue contrast
- Fat/water homogeneity
- Additional Sponsor-Requested Assessments
  - CRF fields (10 blank "Assessment Title" lines with associated 1-5 Likert scales) will be provided on the CRF to accommodate Sponsor-requested elements that may be specified for each MR Procedure Document
    - The investigator is responsible for being aware of any additional elements required by each MR Procedure Docume Mersion number.
    - The investigational site(s) will be notified of any additional instructions for completing comments, and will be responsible for completing the comments field as instructed after appropriate training and instruction has been provided by the Sponsor.

## 6.4. Unexpected Findings

MR scanning in this study is for research purposes only, and is not intended to diagnose or treat any disease or condition. Furthermore, study images shall not be reviewed or provided for diagnostic or any other purposes which may affect patient care. Study images are not being evaluated for specific clinical findings.

However, in the course of performing study procedures in any part of this study (Phase 1 or Phase 2), should the study staff observe unexpected findings, the Principal Investigator may choose to communicate such findings to the subject's parent(s) or legally authorized representative(s) and/or other clinicians involved in the subjects routine clinical care. Are port of an unexpected finding should clearly state that the study MRI scans have been reviewed only for technical purposes as required by the study and are not meant to supplement or replace any clinical MRI exam or MRI report as would be provided for standard of care exams. Further, it should be reported that the study scans were performed on an investigational device which is not yet approved for diagnostic imaging. Thus, any findings described cannot be guaranteed to be accurate or of clinical significance. The study Principal Investigator may note details of what is seen related to the unexpected finding to parent(s) or legally authorized representative(s) and/or, if necessary, to other clinician's involved in the subject's routine clinical care, but no diagnosis should be rendered based on study data. The study Principal Investigator may make recommendations for standard of care imaging follow-up, which, if necessary, will be conducted outside of this study. When an unexpected finding is reported, subjects in this study are then to be managed as patients with regard to standard of care in accordance with the site's policies and procedures.

The Principal Investigator shall complete the study Investigator's Report form regarding unexpected findings, or the noted absence thereof, for every study scan session. The PI may use this form to communicate findings to the responsible clinicians. The form should be stored in the study file, and a copy of the completed form may also be stored in any other location required or recommended by the General Medical Council record keeping guidelines.

Study Number: 114-2014-GES-0035

Protocol: 7.0



## 6.4.1. Follow-up for Unexpected Findings

In Phase 1 of this study, if unexpected findings identified during this study result in referral for further MRI diagnostic evaluation or other medical care according to the standard of care at the investigational site, de-identified images and associated image data from the standard of care MRI may be observationally collected and provided to the Sponsor for engineering development and device optimization purposes. The occurrence of unexpected findings will be reported on the case report form (CRF). This data is being collected for exploratory engineering development and device optimization purposes, to learn more about performance characteristics and potential artefacts in Neonatal MRI scans. Images and associated image data will be provided at the discretion of the Principal Investigator, and may not be available for all patients with unexpected findings.

### 6.5. Withdrawal and Discontinuation Criteria

All subjects must be admitted for care in the NICU or other neonatal or infant care department or unit affiliated with the investigational site at the time of enrolment and scanning to be eligible to participate in this study. If a subject is discharged from clinical care at the investigational site prior to MR scanning, the subject will be withdrawn from the study.

The subject's medical care shall take precedence over any imaging or other procedures associated with the study.

If it is determined during the exam that the study imaging will in any way negatively impact required clinical care, the subject shall be immediately withdrawn from the study.

In the event the subject appears to be in pain or undue discomfort, if potentially destabilizing vital signs are observed by visual inspection or via monitoring equipment, or if the parent(s) or legally authorized representative requests to discontinue study procedures, the study procedures will be discontinued immediately and the subject will be removed from study, as determined necessary by the medically qualified staff at the investigational site. The subject shall be removed from the MR environment as soon as safely possible, and, if necessary, care will be provided to the subject to alleviate any discomfort according to the site's standard of care. Data collected up until the time of withdrawal may still be used and disclosed to the Sponsor for research purposes.

The subject's parent or legal guardian may withdraw him or her from study participation at any time, for any reason without consequence.

The study staff may withdraw a subject at any time for any reason.

The reasons for withdrawal and discontinuation for any subject shall be recorded. These will be reported to the Sponsor.

The EC/IRB should be notified per their notification of subject withdrawal policy. There shall be no negative repercussions to the subject, parent(s) or legally authorized representative, or Study Staff for deciding end any study procedures.

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



# 6.6. Study Flowchart

Table 3– Flowchart detailing the data elements to be collected during each part of the study

| Procedure/<br>Data Element | General Procedures (time interval) | Recruitment<br>/<br>Screening | Pre-Scan | MR<br>Scanning | Post-Scan | Reader/<br>Evaluator<br>Assessments |
|---|---|---|---|---|---|---|
| Quality Control Scan | Sponsor-set interval(s) <sup>1</sup> | | | | | |
| Specific Absorption Rate | | | | X | | |
| (SAR) Scans | | | | | | |
| Running MR Scan | Daily | | | X | | |
| Session Log | verification | | | | | |
| MR Procedure | Prior to | | | | | |
| Documents | enrolling first | | | | | |
| (Prepared by Sponsor) | subject, | | | | | |
| | thereafter at | | | | | |
| | Sponsor-set | | | | | |
| | regular | | | | | |
| | interva l <sup>1</sup> | | | | | |
| Qualitative Investigator | Within ∼3 | | | | X | |
| Summary | business | | | | | |
| (Prepared by PI) | days of | | | | | |
| | completing | | | | | |
| | MR | | | | | |
| | Procedure | | | | | |
| | document | | | | | |
| Inclusion/Exclusion | activities | X | | | | |
| Collect subject | | Λ | X | X | X | |
| Information | | | Λ | Λ | Λ | |
| MR Safety | | X | X | X | X | |
| (subject and any persons | | 71 | 71 | 21 | 71 | |
| accompanying him or | | | | | | |
| her into scan room) | | | | | | |
| Application/Removal of | | | X | | X | |
| Swaddling (if | | | | | | |
| used)/Padding | | | | | | |
| Transport | | | X | | X | |
| Environmental | | | X<br>X | | X<br>X | |
| conditions | | | | | | |
| MR Procedure | | | | X | | |
| Document Identification | | | | | | |
| (Version number) | | | | | | |
| MR Scanning | | | | X | | |
| Information | | | | | | |
| Software/Hardware | | | | X | | |
| components used | | | | (Phase 1 only) <sup>2</sup> | | |
| MR Scanner Technical | | | | X | | |
| Issues/Malfunctions | | | | | | |
| Additional Sponsor- | | | X | X | X | X(reader only) |
| Requested Assessments | | | | | | |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Procedure/<br>Data Element | General<br>Procedures | Recruitment / | Pre-Scan | MR<br>Scanning | Post-Scan | Reader/<br>Evaluator |
|---|---|---|---|---|---|---|
| | (time interval) | Screening | (1 6 1: | (1.6.1 | (1.6. 1: 16. | Assessments |
| | | | (defined in MR | (defined in MR | (defined in MR<br>Procedure Doc) | (defined in MR<br>Procedure Doc) |
| | | | Procedure | Procedur | Procedure Doc) | Flocedule Doc) |
| | | | Doc) | e Doc) | | |
| MR Images and Data | | | | X | X | X |
| 8.2.2.2. | | | | | | (access to) |
| Evaluable | | | | | | X |
| (Diagnostic) Non- | | | | | | (reader and |
| evaluable (Non- | | | | | | evaluators) |
| diagnostic) Assessment | | | | | | |
| Image Quality | | | | | | X |
| Assessments | | | | | | (reader only) |
| Overall image quality | | | | | | X |
| (based on | | | | | | (reader only) |
| investigator's | | | | | | |
| experience | | | | | | |
| Image contrast | | | | | | (" |
| Presence ofartefacts | | | | | | (reader only) |
| Presence oartelacts | | | | | | / ` ` |
| Signal to noise ratio | | | | | | (reader only)<br>X |
| (SNR) | | | | | | (reader only) |
| Tissue contrast | | | | | | (reader only) |
| rissue contrast | | | | | | (reader only) |
| Fat/water separation | | | | | | X |
| | | | | | | (reader only) |
| AEs/SAEs | | | Х | X | Χ | , , , , , |
| | | | (From | | (to removal | |
| | | | placemen | | from | |
| | | | t on | | swaddle/paddin | |
| | | | swaddle, | | g and return to | |
| | | | if used, or | | clinical care | |
| | | | if not used | | environment) | |
| | | | from | | | |
| | | | removal | | | |
| | | | from | | | |
| | | | clinical | | | |
| | | | care | | | |
| | | | environm | | | |
| MR System | | | ent to MR) | Х | | |
| Errors/Issues | | | | ^ | | |
| MR | | | X | Х | Х | |
| Component/Accessori | | | | | | |
| es Errors/Issues | | | | | | |
| Usability Assessments | | | | | | |
| SystemUsability Scale | Operator | | | | | |
| (SUS) | completes at | | | | | |
| , , | end-of- | | | | | |
| | scanning for | | | | | |

Study Number: 114-2014-GES-0035

Protocol: 7.0



| Procedure/<br>Data Element | General<br>Procedures<br>(time interval) | Recruitment / Screening | Pre-Scan | MR<br>Scanning | Post-Scan | Reader/<br>Evaluator<br>Assessments |
|---|---|---|---|---|---|---|
| | each MR Procedure Docin Phase 1 and at end | · · | | | | |
| | of Phase 2 | | | | | |
| User Experience Scale (UXS) | Operator<br>completes<br>end-of-<br>scanning for<br>each <i>MR</i><br><i>Procedure</i><br><i>Doc</i> in Phase<br>1 and at end<br>of Phase 2 | | | | | |
| Usability for Device | | | | | Х | |
| Components | | | | | | |
| Qualitative Investigator<br>Summary | PI or<br>designee<br>completes<br>for each<br>Sponsor<br>Investigator<br>meeting in<br>Phase 1 | | | | | |
| End-of-Phase Summary<br>Report | PI or<br>designee<br>completes at<br>end of Phase<br>1 and Phase<br>2 | | | | | |

*Note*: X = tobe conducted in indicated part of the study

- 1. Conducted at intervals set and determined by the study Sponsor. The PI rates complete additional general quality scans that do not use human subjects (i.e. phantonat) any time during the study
- For Phase 1scanning only; In Phase 2 these components are fixed all subjects by the applicable MR
   Procedure Document ersion

## 7. TRAINING PLAN

# 7.1. Training Plan for ResearchDevice/Product

Study Staff will be trained on the use of device system, its components, and Sponsor-provided accessories such as the Sponsor-provided patient monitoring equipment. The Sponsor will provide initial instructions for use of the device and swaddles and, as necessary, subsequent training on any changes to the device, including any necessary storage and handling requirements, preparation for use, any pre-scan checks of safety and performance and any precautions to be taken after use, (e.g. disposal).

No training will be conducted on human subjects.

Study Number: 114-2014-GES-0035

Protocol: 7.0



#### 7.1.1. MR Procedure Documents

The PI is responsible for ensuring that all MR scan operators that will be operating the research device will be made aware of and, if necessary, provided training on scanning proceduresat the beginning of the study and after any new version of the Procedure Document is released by the Sponsor to the investigational site

## 7.1.2. Configuration Changes

The PI is responsible for ensuring that all Mean operators that will be operating the research device will be made aware of and, if necessary, provided training on device configuration changes released by the Sponsor to the investigational site.

## 7.2. Training Plan for Protocol

Study staff will be trained on the Study protocol and Study procedures, including completion of Informed Consent Forms (ICFs), Case Report Forms (QRR 4), ocedure Documes, and other study documentation

Trainingwill also be provided to ensure appropriate storage and handling of images and data. All study staff will be required to be trained @ood Clinical Practic(GCP) guidelines per ISO 141552011.

A record of all formal training attendance and date conducted will be stored in the Site Regulatory Binder and provided to the Sponsor for inclusion in the Sponsor's Clinical History File (CHF).

#### 8. DATA ANALYSISNDSTATISTICS

# 8.1. Statistical Analysis Methods

#### 8.1.1. Sample Size Determination

Based on the literature, studies including lewirth weight neonates commonly assume a 20% dropout rate<sup>28</sup> Compared to gold standard, approximately 82% of images attained from neonates/infants with MRI are diagnosticallyseful (evaluable)in part due to subject movement during scanning<sup>29</sup> Theenrolment quota calls for 30 (Phase 1) an (Phase 2) evaluable image sets. More than one image set may be collected from a single subject; however, this case is exceptional and may not be common.

This study requires a population of such as that:

$$0.82N - (0.82 \times N)(0.2) = (30 \text{ phase } 1 + 5 \text{ phase } 2)$$

To satisfy this requirement, a minimum population size *M*=53 is required. This is approximated upwards to *M*=60 to account for unforeseen contributions to dropout or evaluable image rates in sensitive neonate and infapopulations. It is prospectively expected that Phase 1 of this study may be ended early if required data for engineering purposes is collected before the maximum number of subjects enrolled; it is also prospectively expected that Phase 2 of this studyay be ended early if required data for regulatory submission is collected before the maximum number of subjects are enrolled in this Phase. Any determination to end the study before the expected number of subjects has been enrolled will be provided by th Sponsor, in writing, to the investigational site.

Study Number: 114-2014-GES-0035

Protocol: 7.0



### 8.1.2. Statistical Analysis Methods

As necessary to support regulatory submission, continuous variables will be summarized with standard descriptive statistics including counts, means, standard deviations, medians, and minimum, maximum. Categorical variables will be summarized with frequencies and percentages.

## 8.1.3. Other Analysis Methods

Images and associated data being collected in this study are intended for use on a persubject basis for engineering purposes.

Upon completion of this study, the Sponsor's authorized research and engineering program may utilize data collected in this study in full or in part for authorized engineering purposes. The principal investigator (PI) at each site may be asked to provide electronically tabulated data summaries for subject demographics and other descriptive data summarizing study results. PI-prepared data tabulations will not be controlled or verified by the Sponsor. These results are collected for learning purposes only, and any PI-provided data tabulations will be summarized in the final study report for reference only. Any direct or derived results from PI-prepared data tabulations will not be used by the Sponsor for regulatory submissions.

## 8.2. Interim Analysis

There are no interim cohort-based statistical analyses for this study. At the Sponsor's discretion and per local EC/IRB requirements, the status of enrolment and other subject data may be summarized at any time determined by the Sponsor during this study.

## 8.3. Handling of Missing Data

The Sponsor may descriptively summarize the primary performance and safety endpoints from Phase 1 and Phase 2 of this study, including the descriptive statistical summary of patients that exhibit a body temperature rise of more than  $0.5\,^{\circ}$ C from acclimated prescanning baseline body temperature (resulting in an Expression Monitor alarm during scanning). If the Sponsor observed that the dataset for any subject is incomplete, additional clarification from the investigator may be requested. The Sponsor may additionally request copies of any clinical imaging datasets (including MRI scan datasets and other clinically indicated imaging examinations) that are conducted as follow-up to unexpected findings observed in this study.

## 8.4. Pass/Fail Crteria of the Study

The study will be considered successful if sufficient evidence is collected to inform the performance and safety of the 3.0T Neonatal MRI investigational device in a representative population of neonates and/or infants, in accordance with Annex Xof the European Medical Device Regulation.

Study Number: 114-2014-GES-0035

Protocol: 7.0



# 9. OTHER INTERIM ACTINES (QUALITATIVE INTENRISUMMARIES)

## 9.1. Phase 1Qualitative Investigator Summary

For Phase 1 of this study, the PI is responsible for preparing qualitative Interim Summaries based on meetings between the Sponsor and investigator, as described in <u>Section 9.1. Phase 1 Qualitative Investigator Summary</u> (Phase 1 only).

These documents, along with images and data collected to date, will provide a basis for the Sponsor's determination of MR Procedure Document

## 9.2. Phase 1 and Phase 2 End-of-PhaseInterim Reports

A total of two Endof-Phase Interim Reports will be prepared by PI at the end of enrolment for Phase 1 and the end of enrolment for Phase 2. The PI widescriptively summarize the subject population and imaging results collected to date his may include data tabulations, at the discretion of the PThe Phase 1 Endof-Phase Interim Report may be considered by the Sponsor idecision-making activities required for Phase 2, and may be summarized in the Sponsor's final clinical study report-prepared data tabulations will not be controlled or verified the Sponsor results are collected for learning purposes only, and any Pprovided data tabulations will be summarized in the final study report for reference only. Any direct or derived results from Prepared data tabulations will not be used by the Sponsor for regulatory submissions.

#### 10. DEVIATIONS

## 10.1. Management of Protocol Deviations

All human MR scanning with the investigational device used in this study must be conducted under a current MR Procedure Documentersion. If any clinical scan procede is conducted that is not compliant with the current MR Procedure Documentersion it will be considered a deviation and should be reported according to the following guidelines

Deviations to the protocol may occur when necessary to protect the lifeponysical well-being of a subject

Except in an emergency, prior approval by the ponsoris required for changes in planned deviations from this protocol

If these changes affect the scientific soundness or the safety and welfare of the subject, prior ECIRBapproval is also required

Planned Protocol Deviation documentation must be filed in the Site Study Regulatory Binder

There are two types of unplanned protocol deviations, critical deviations and roritical deviations

All deviations must be documented and reported, the criticality of the deviation will determine the reporting path

#### **Critical Deviations:**

Deviations that significantly affect the safety, efficacy, integrity or conduct of the study

Study Number: 114-2014-GES-0035

Protocol: 7.0



These deviations must be reported to the Sponsor no later than 5 working days from awareness of occurrence and reported to the EC/IRB per the deviation reporting policy.

If an Investigator uses a device without obtaining informed consent, the Investigator shall consider this a critical deviation and report the event to the Sponsor and the EC/IRB within 5 working days of the occurrence.

#### Non-Critical Deviations:

Protocol deviations that DO NOT significantly affect the safety, efficacy, integrity or conduct of the trial.

These deviations must be documented on the Case Report Form Protocol Deviation page and will be reviewed by the study monitor.

#### 11. COMPLAINT HANDLINGNDADVERSE EVENT REPTORS

## 11.1. Foreseeable Adverse Events an Device Effects

MRI is generally considered safe for adults and babies because it does not involve exposure to ionizing radiation, such as x-rays. MRI of 4T or less is considered non-significant risk for infants and neonates, and population-specific risks are well described. <sup>26,30,31,32,33,34,35</sup> The known risks typically associated with 3TMRI scans in this study are listed below and have been mitigated by the Sponsor to levels that are as low as reasonably practicable (ALARP), to levels equivalent or less than MRI using commercially released scanners:

*Movement of Metal Objects* Magnetic fields in MRI can cause internal or external ferrous metal (e.g. implants, umbilical cord clamps, oxygen tanks, infant security bands, scissors, paperclips, and pens) small enough to be innocuous to adults to move or become projectile, leading tominor injuries like cuts/bruises and, in rare cases, serious injury or death.

Thermal Effects: Body temperature can change due tenvironmental cooling and/or MRI radiofrequency (RF) warming. Typicalexific absorption rates(SAR) during study MRI scanning are not expected to cause injury. In rare cases, serious burns can occur that are typically related metallic object presence or improper patient positioning.

Semi-permanent Cable/Device RemovalChest leads and other semipermanent attached cables/devices can warm and electronics can function abnormally, potentially causing discomfort, injury, interruption of care, and, in rare cases, serious destabilization. Devices not known to be safe in the MRI environment may be removed or replaced when doing soldwo not detrimentally impact normal medical care, otherwise the subject will bethdrawn.

Peripheral Nerve Stimulation: Transient skin sensations ('tingling') or peripheral nerve stimulation (PNS) is related ttB/dt and gradient rise time, and iexpected to berare in neonates and infants due to small skin surface area and conservative device thresholds. Subjecting infants to sudden, rapidly changing gradient magnetic fields during imaging can, induce circulating currents in conductive tissues of the body that typically are not painful and resolvespontaneously though, in theory, discomfort or pain from IPS in infants is possible.

Acoustic Noise. High noise levels in the scan room and in the bore of the scannel wring MRI scanning may cause discomfort but are notormally hazardous with proper heaing protection. Spontaneously resolving hearing loss initus typically related tomproper hearing protection can, in rare cases, become chronic or severe. Hearing protection

Study Number: 114-2014-GES-0035

Protocol: 7.0



(combination of earplugs or ear plugs combined with earmuffs to achieve noise reduction of ≥22dB is mandatory during MRI in this study)

Adverse Effects due tdDelay of care Though discontinuation of study procedures for urgent medical care is not anticipated, unexpected regent care may be delayed due to removal from the MRI on other study devices. The expected delay is only a few minutes, but there is a risk that any amount of delay could detrimentally impact urgent medical care.

In addition, there are possible, but not anticipated risks that have been identified for the Neonatal MRI deviceduring development. These risks have be interested and mitigated to levels ALARBy the Sponsor and are described as follows:

Airflow Interruption: In rare cases, blockage of the bore of timevestigational 3.0 Theonatal MRIdevice, particularly at the head end of the scanner, can cause interruption of normal airflow in the bore of the scanner. Through proper measurement of the subject, combined with visual inspection of the bore of the scanner once the subject is placed in the scanner the scan operator will ensure that no blockage of the bore of the MR scanner exists.

**Swaddlerisk**: Compression by the swaddle can cause discomfort and, in rare casses serious injury usually due tostudy procedures not being followed.

**Fall.** During transport or scanning, infants and neonates may be at increased risk of fall from the height of the MRI table or transport devices, typically due to improper use. The risk of fall is not expected to be greater than in routine transport and the height of all device components complies with regulatory requirements.

Like routine MRI scanning of <4.0 MRI procedures conducted with the 0.0 Theonatal MRI investigational device rarely cause harm when performed a directed by trained staffusing appropriate procedures as described in this protocollevice documentation and in Sponsor provided training The risks of AEs and SAEs been mitigated by the Sponsor the vels ALARP. If the Sponsor learns any new information that would increase to is study, the PI will be notified in writing.

#### 11.2. Adverse Event Definitions

Adverse Event (AE) as defined by EN ISO 14155-2011: any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device.

Serious Adverse Event (SAE)s defined by EN ISO 14155 – 2011: an adverse event that

- (a) led to death;
- (b) led to a serious deterioration in the health of the subject, that either resulted in:
  - (1) a life-threatening illness or injury, or
  - (2) a permanent impairment of a body structure or a body function, or
  - (3) in-patient or prolonged hospitalization, or
  - (4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to body structure or a body function;

Study Number: 114-2014-GES-0035

Protocol: 7.0



(c) led to fetal distress, fetal death or a congenital abnormality or birth defect.

**Anticipated:** Any adverse event and/or reaction, the specificity or severity of which is consistent with the EC/IRB approved informed consent, protocol, investigator brochure, or product labelling.

**Unanticipated adverse Device effect**: Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.

## 11.3. Management of Adverse Event Reporting

Any adverse events will be recorded in the subjects study record and the Adverse Event Case Report Form. The following information should be obtained:

- Description of Event
- Date of onset and resolution
- Intensity (mild, moderate, severe)
  - <u>Mild</u>: Symptom(s) barely noticeable to the subject or does not make the subject uncomfortable. The AE does not influence performance or functioning. Prescription drugs are not ordinarily needed for relief of symptom(s).
  - Moderate: Symptom(s) of a sufficient severity to make the subject uncomfortable.
     Performance of daily activities is influenced. Treatment of symptom(s) may be needed.
  - **Severe** Symptom(s) of a sufficient severity to cause the subject severe discomfort. Treatment for symptom(s) may be given.
- Serious (yes/no)
- Relationship to device (unrelated, possibly related, probably related)
  - Unrelated: The adverse event is reasonably expected to be related to (or caused by) a
    concurrent illness, effect of another device/drug or other cause, and is unlikely
    related to the investigational product
  - <u>Possibly related</u> The adverse event is reasonably expected to be related to the investigational product, and an alternative actiology is equally or less likely compared to the potential relationship to investigational product
  - <u>Probably related</u>: There is a strong relationship to investigational product, or recurs on re-challenge, and another aetiology is unlikely, or there is no other reasonable medical explanation for the event.
- Treatment given and/or action taken (procedure stopped, withdrawn from study, no action)
- Anticipated (yes/no)

Adverse events that occur during a subject's active enrolment (as described in Section 6.3.1. - Pre-MR Scanning Activities: Duration of Active Enrolment) will be reported to the local EC/IRB per their policy and, if applicable, to regulatory agencies. Medical events that occur outside of

Study Number: 114-2014-GES-0035

Protocol: 7.0



the active study during observational data collection, such as during standard of care followup conducted for any unexpected findings, will not be considered study adverse events.

# 11.4. Management of Serious Adverse Evenand Unanticipated Adverse Device Effect Reporting

All SAEs and or UADEs will be documented as above and reported in writing to the Sponsor within 72 hours of knowledge of the event The Investigator shall submit the Adverse Event Case Report Form and GEHC\_GQP\_10.07.005\_F002 Site Notification and Assessment of Serious and Unexpected Adverse Events (DOC0910335) with redacted supporting documentation to SAE mailbox.

If the event resulted in the death of a subject, the event shall also be reported via telephone to the Sponsor within 24 hours of knowledge of the event. SAEs will be reported to the local EC/IRB per their policy and, if applicable, to regulatory authorities in accordance with their requirements.

#### Sponsorcontact for SAEsand/or UADEs

Jeff Hersh MD +1-262-366-7295 Fax 800-888-3983 E-mail: SAE@geom

If additional information (e. outcome of event, datevent resolved, additional treatments) is required to submit a followup report, the Investigator shall update the AE CRF and resubmit to Clinical Affairs

The Investigator shall submit the followip SAE and/or UADE report to the local/ECBper their policy.

# 11.5. Management of Device Complaints

Any complaints regarding the operation of the eviceor software or any malfunctions are to be reported to the Clinical Affair Project Manager

#### Sponsorcontact for Device complaints:

Yvonne CelestialClinical Affars Project Manager *Phone*+33 130709133 *Email* MarieYvonne.CELESTIAL@ge.com

## 12. EARLY TERMINATION ORSPENSION

# 12.1. Criteria for Early Termination or Suspension

The study may be terminated early if the ponsordetermines that unanticipated adverse event(s) presents an unreasonable risk to subjects or for any other reaso passnsor determines to be appropriate

Study Number: 114-2014-GES-0035

Protocol: 7.0



The Phase 1 Interim Report will be used by the Sponsor to determine if Phase 2 should be conducted and which version(s) of the *MR Procedure Document* ll be applied in Phase 2 Consistent MR procedures will be used for all subjects throughout Phase 2.

Termination shall occur no later than 5 working days after the one of the determination and no later than 15 working days afte Sponsorfirst received notice of the effect.

The Sponsorwill promptly notify the Investigators of any determination to terminate the study outside of the protocol timeframe

The Sponsorwill provide each Investigator with written guidelines/instructions on termination processes and timelines

The Investigator is responsible for reporting the early termination to their local ALROB

In the event of early termination after Phase 1, the Investigator remains responsible completing a descriptive report of the results

## 12.2. Withdrawal of EC Approval

The Investigator is to notify the Sponsor of any withdrawal of EC/IRB approval within 5 working days of such occurrence.

If the EC/IRB terminates or suspends its approval of the Study, the Investigator will promptly notify Sponsor and provide a detailed written explanation of the termination or suspension.

Upon receipt, the Sponsor will provide written guidelines/instructions on subject withdrawal/termination processes and timelines.

# 13. ETHICS COMMITTEE MODREGULATORY FILINGS

# 13.1. Regulatory Authority Approval Requirements (Global)

In the United Kingdom (UK) the use of the device is subject to regulation by the Medicines and Healthcare Products Regulatory Agency (MHRA), in compliance with the European Medical Device Directive 93/42/EEC. MHRA authorization is required prior to enrolling subjects. The Sponsor will notify the PI in writing to authorize subject enrolment.

# 13.2. Ethics Committee Approval Requirements

This study is to be submitted to the EC/IRB for review and approval prior to enrolling subjects.

The Investigator is responsible for keeping approval current and maintaining appropriate correspondence and reports.

Copies of all EC/IRB applications, approval letters, Informed Consent Forms (ICF) and other correspondence are to be sent to the Sponsor, with originals kept in the Site Study Regulatory Binder.

# 13.3. Management of Protocol Revisions/Amendments

All protocol amendments will be approved and released by the Sponsor.

Study Number: 114-2014-GES-0035

Protocol: 7.0



## 13.4. Informed Consentand Privacy Requirements

Per European Medical Device Directive 93/42/EEC, the following will be required for all neonate/infant subjects enrolled in this study:

- a. The parent(s), or guardian(s), or legally authorized representative(s) will be required to sign the informed consent form;
- b. If it is the determination of the EC/IRB that both parent(s) or guardian(s) sign the informed consent form, that will occur except in the case of deceased, unknown, incompetent, or not reasonably available parties, or when only one parent has legal responsibility for the care and custody of the child if consistent with (EU) law and any other applicable laws and/or regulations at the site where the study is being conducted.
- c. Permission by parents or legally authorized representative will be documented in accordance with, and to the extent required, by ISO 14155: 2011 (EU).

Informed consent will be documented in each subject file.

The Investigator or designee will consent the subject's parent(s), or guardian(s), or legally authorized representative(s) per regulatory guidelines, which includes the right to have ample time to review the ICF and have all questions answered to their satisfaction. Subjects may sign the ICF at the time it is presented if all of his/her questions have been answered. In the event that a the parent(s), or guardian(s), or legally authorized representative(s) require additional time or wishes to discuss the ICF with others, he/she will be allowed to take the ICF home prior to signing to review with family members or others before making a decision.

The parent(s), or guardian(s), or legally authorized representative(s); the person who consented the subject; and the investigator must sign and date the ICF document prior to a subject being included in the study.

The subject's parent(s), or guardian(s), or legally authorized representative(s) will be given a copy of the signed informed consent form and the original will be retained with subject files.

#### 13.4.1.Consent for International Transfer and Use of Deidentified Data

The informed consent form (ICF) will explain that some data collected as part of this study may be transferred outside of the European Union (EU), including to the United States (US) and to other countries which may not provide the same level of data protections as the EU. Steps will be taken in order to protect the confidentiality of the data subjects. Applicable local laws and regulations for the transfer and use of clinical study data will be followed.

## 14. DATAANDQUALITY MANAGEMENT

# 14.1. Management of Data

Images and data will be collected from subjects enrolled in this study and pseudonymised using subject identification designation (SID). The resulting data will be key-coded and will not contain any direct identifiable personal information (e.g. no name).

GE Healthcare and authorized representatives may use image and associated data from this study for future technology development, marketing purposes, publications, regulatory use or

Study Number: 114-2014-GES-0035

Protocol: 7.0



any other possible use. The images and associated image data collected from unexpected findings may be used for engineering development and device optimization purposes. Phase 2 data is collected with the intent of use in regulatory submissions, such as CE mark.

The approved Data Management Plan (DMP) will be located in the study's clinical history file maintained by the Sponsor.

#### 14.1.1.International Transfer and Use of Deidentified Data

In the case where personal data is transferred outside of the European Union (EU), it will be transferred to the United States (US) and other countries which may not provide the same level of data protections as the EU. Steps will be taken in order to protect the confidentiality of the data subjects. Applicable local laws and regulations for the transfer and use of clinical study data will be followed.

## 14.2. Subject Deidentification

Not Applicable This section is not applicable for studies conducted in this region and is superseded by Section 13.3 Subject Pseudonymisation.

## 14.3. Subject Pseudonymisation

All subject data that is submitted to the Sponsor will be identified by the use of a unique subject number assigned as midentification code to the Subject, without delentification. The scan operator will enter the identification number in the system complete pseudonymisation

The assigned subject identification numbercoording to the Sponsor's Data Management Plan DMP).

Each participating site will maintain a subject identification log, which is a list of all subjects who are enrolled in the study, along with their address and medical record number in the event that they must be contacted in the future

The Sponsor will not receive a copy of the subject identification log

## 14.4. Completion of Case Report Forms (CRFs)

Data will be collected using paper CRFs, and data file transfers

GEHC will provide CRFs and the instructions for their completion.

To ensure the quality and integrity of the data, it is the responsibility of Priencipal Investigator or designee in a timely mannet complete a CRF for each subject who is enrolled to participate in this studyCRFs will be completed as information bomes available.

If errors or omissions are found in the course of a CRF audit, or data review. Who to File (NTF) or Data Clarification Form (DATF) be generated and the error, omissions or clarifications will be corrected on these forms

The Principal Investigator will sign and datelte indicated places on the CRF

The Principal Investigator's signature will indicate that a thorough inspection of the data has been made and will thereby certify the contents of the form

Study Number: 114-2014-GES-0035

Protocol: 7.0



#### 14.5. Record Retention at the Stie

All records pertaining to the conduct of the study, including Case Report Forms, Informed Consent Forms, Ethics Committee correspondence, and other study documentation must be retained at the Site for inspection at any time by the GEHC Study Monitor or designee. These records will be maintained according to GEHC Retention Policies. Elements should include the following:

- Subject Files containing the completed subject CRFs
- Regulatory Binder containing the protocol and amendments, EC/IRB submissions and approvals, (blank and signed/dated) Informed Consent Form(s), and Site study logs
- Reference Manuals containing the resource list, responsibilities of the Investigator, Sponsor, adverse event and informed consent guidelines, study aids (training material, device screen shots), and central supplier instructions.

No records will be destroyed without GE Healthcare notification and approval.

### 15. MONITORING PLAN

## 15.1. Brief Description

In collaboration with the site, the Sponsor will ensure proper monitoring of the study to confirm that all the clinical requirements are met. Monitoring visits will ensure adherence to the protocol, completion of informed consents, EC/IRB review of the study, maintenance of records, primary outcomes review and review of the CRFs and source documentation for accuracy and completeness.

# 15.2. Reference to Approved Monitoring Plan

The approved monitoring plan will be located in the study's clinical history file (CHF) maintained by the Sponsor.

#### 16. PUBLICATION FLOCY

The Sponsor and its authorized representative may also utilize the images and data, in a fully anonymized format, for scientific publication(s), presentation(s) at scientific meetings or trade shows, product development, marketing materials, educational and training, support of global regulatory submissions, or other purposes authorized by the Sponsor in accordance with applicable laws and regulations.

Publications by investigators, study staff, and others involved with the study and/or investigational site will be governed by the contractual agreement between the Sponsor and site.

#### 17. ADDITIONAL COUNTRSPECIFIC REGULATORS OR JIREMENTS

Applicable regulations in the UK will be followed in this study.

Study Number: 114-2014-GES-0035

Protocol: 7.0



#### 17. REFERENCES

- 1. US FDAGuidance for Industry and FDA Staff: Premarket Assessment of Pediatric Medical D May 14, 2004.
- 2. Malik S, Beqiri A, Price A, Teixeira J, Hand J, Hajnal J. Specific absorption rate in neonates undergoing magnetic resonance procedures at 1.5 Tand 3 T. *NMR Biomed* 2015;28(3):344-52.
- 3. Glass H, Bonifacio S, Sullivan J, et al. MRI and Ultrasound Injury in Preterm Infants with Seizures. *J Child Neurol*2009;24(9):1105-1111.
- 4. Arthur R. Magnetic Resonance Imaging in Preterm Infants. *Pediatr Radio*: 593–607.
- 5. Barkovich A. R Imaging of the Neonatal Brain. Neuroimaging Clin. N. Am. 2006;16:117–35–viii–ix. *Neuroimaging Clin N Am 2008*006;16:117–35–viii–ix.
- 6. Arthurs O, Edwards A, Austin T, Graves M, Lomas D. The challenges of neonatal magnetic resonance imaging. *Pediatr Radiol*2012;42(10):1183-94.
- 7. Oishi K, Faria A, Mori S. Advanced Neonatal Neuro MRI. *Magn Reson Imaging Clin N Am* 2012;20:81–91.
- 8. Rutherford M, Biarge M, Allsop R. MRI of perinatal brain injury. *Pedatr Radiol*2010;40:819–833.
- 9. Tkach J, Hillman N, Jobe A, et al. An MRI system for imaging neonates in the NICU: initial feasibility study. *Pediatr Radiol*2012;42(11):1347-56.
- 10. Ment LR BHBPea. Practice parameter: Neuroimaging of the neonate: Report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. *Neurology* 2002;58:1726–1738.
- 11. Kilian A, Schaible T, Hofmann V. Congenital diaphragmatic hernia: Predictive value of MRI relative lung-tohead ration compared with MRI fetal lung volume and sonographic lung-to-head ratio. *AJR*192:153–158.
- 12. Dumoulin C, Rohling K, Piel J, et al. Magnetic Resonance Imaging Compatible Neonate Incubator. *Concepts in Magnetic Resonance 2002;15:41128*. 2002;15:117–128.
- 13. Whitby E, Griffiths P, Lonneker-Lammers T, et al. Ultrafast Magnetic Resonance Imaging of the Neonate in a Magnetic Resonance-Compatible Incubator with a Built-in Coil. *Pediatrics* 2004;113:e150–2.
- 14. Blüml S, Friedlich P, Erberich S, Wood J, Seri I, Nelson M. MR Imaging of Newborns by Using an MR-Compatible Incubator with Integrated Radiofrequency Coils: Initial Experience. *Radiology* 2004;231(594–601).
- 15. Rutherford M. MRI of the neonatal brain. *Saunders, UK*2001. Available at: http://www.mrineonatalbrain.com.
- 16. Tkach J, Hillman N, Jobe A, Loew W, Pratt R. An MRI system for imaging neonates in the NICU: initial feasibility study. *Pediatr Radiol*2012;42(11):1347-56.
- 17. Barkovich A, Kjos B, Jackson D, Norman D. Normal Maturation of the Neonatal and Infant Brain: MR Imaging at 1.5 T. *Radiology 1988*;166:173–180.
- 18. Johnson M, Pennock J, Bydder G, Dubowitz L, Thomas D, Young I. Serial MR Imaging in Neonatal Cerebral Injury. *Am J Neuroradiol* 987;8:83-92.
- 19. McArdle C, Richardson C, Nicholas D, Mirfakhraee M, Hayden C, Amparo E. Developmental Features of the Neonatal Brain: MR Imaging Part I. Gray-White Matter Differentiation and Myelination. *Radiology* 1987,162:223–229.

Study Number: 114-2014-GES-0035

Protocol: 7.0



- 20. Dumoulin C, Rohling K, Piel J, et al. Magnetic Resonance Imaging Compatible Neonate Incubator. *oncepts in Magnetic Resonanc***2**002;15:117128.
- 21. Stokowski L. Ensuring safety for infants undergoing magnetic resonance imaging Neonatal Care 2005;5(1):1427.
- 22. Plaisier A, Raets M, van der Starre C, et al. Safety of routine early MRI in preterm in *Radiatr* Radiol 2012;42(10):120**5**1.
- 23. BenaventeFernández I, LubiárLópez P, Zuazojeda M, JiménezGómez G, Lechugsancho A. Safety of magnetic resonance imaging in preterm infantacta Paediatr 2010;99(6):853.
- 24. Chaves A, Cava J, Simpson P, Hoffman G, Samyn M. Infant cardiac magnetic resonance in using oscillatory ventilation: safe and effective ediatr Cardiol 2013;34(5):1205.
- 25. Blüml S, Wisnowski J, Nelson M, Paquette L, Panigrahy A. Metabolic **Matural** White Matter Is Altered in Preterm Infants*PLoS One*2014;9(1):e85829.
- 26. Stokowski L. Ensuring Safety for Infants Undergoing Magnetic Resonance Ima**tileg**/scape *Multispecialty: Advances in Neonatial Ca*2005;5(1):1427.
- 27. Schenck J. Safetof Strong, Static Magnetic Fields Mag Res Imq2000;12:219.
- 28. Alibadi F, Askary R. Effects of TaetKenesthetic Stimulation on Low Birth Weight Neonatesan *J Pediatr* 2013;23(3):289294.
- 29. Anbeek P, Vincken K, Groenendaal F, Koeman A, Osarh M, van der Grond J. Probabilistic bratissue segmentation in neonatal magnetic resonance imagin@ediatr Res2008;63(2):1583.
- 30. Maalouf E, Counsell S. Imaging the preterm infant: practical issuatherford MA, ed. MRI of the Neonatal Brain London, England: WB Saunders; 2002.
- 31. Groenendaal F, Leusink C, Nijenhuis M, Janssen M. Neonatal life support during magnetic resonance imaging *J Med Engin Techno* 2002;26:7474.
- 32. ECRI*Hazard report: patient death illustrates the importance offnering to safety precautions in magnetic resonance environmen***2**904.
- 33. Shellock F. Magnetic resonance safety update 2002: implants and devided agn Reson Imaging 2002;16:485496.
- 34. Formica D, Silvestri S. Biological effects of exposure to metignresonance imaging: an overview. *BiolMedical Engineering OnLin*2004;3(11).
- 35. McJury M, Shellock F. Auditory noise associated with MR procedures: a reviewagn Reson Imaging 2000;12:3745.

Study Number: 114-2014-GES-0035

Protocol: 7.0



| APPENDIX A EXAMPLE OF | VESTIGATOSUMMARYDOCUMENT |
|---|---|
| ThisInvestigator Summaryvill be complete<br>the SponsorInvestigator meeting conduct | ed by thePlor delegatewithin approximatelythree β)days of |
| the Sponsoninvestigator meeting conduct | Date (DD/Mmm/YYYY) Start Timend Time |
| SummaryNumber | Applicable MR Procedure Docume Mersion: |
| Subject Numbers lecord subjects that con | nplete <b>t</b> heseproceduræ): |
| Comments on current workflow, usability additional pages, if necessaly, | , scanning per MRocedure Document listed abovea(tach |
| Sample Docur | ment-Not for Study Use |
| (Please usenos | t current Sponsorprovided |
| doc | ument version) |
| Comments/Suggestions for future Workfl pages, if necessaly | ow, Usability, Scanning and Apprtimization (attach additional |
| Signature of Principal Investigator deleg | ate Date Completed |
| Printed Name of Principal Investigatour d | elegate |
| Signature of Clinical Affairs Project Manag | ger Date Received by Sponsor |
| Printed Name of Sponsor Representative | <del></del> |

Please submit the completed Investigator Summary within approximately <u>3 business days</u> of each completing the activities described in the current MR *Procedure Document* Submit to:

Yvonne Celestial, Clinic Affairs Project Manager Phone +33 130709133 Email Marie Yvonne. CELESTIAL@ge.com

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| APPENDIX BEXAMPLE OF PROCEDURE DOCUMEN | |
|---|---|
| The Sponsor provided this MR Procedure docu | The Sponsor provided this MR Procedure document on Date (DD/Mmm/YYYY) |
| MR Procedure DocumeNtersion Effective | |
| | Date |
| (DD/Mmm/YYYY) Specific Instructions for procedures to be performance. | me@attach additional pages, if necessary |
| Sample Document-Not for Study Use | |
| (Please usenost current Sponsorprovided | |
| documentversion) | |
| SponsorRequested Assessments of performance on a51Likert Scale mark each assessment required | |
| ☑ Overall Image Qualit <b>/required for all subjects)</b> | Other Assessments: |
| Other Engineering Performance Measures | (specify) |
| Performance parametersp(ecify) | (specify) |
| Performance parametersp(ecify) | (specify) |
| Performance parametersp(ecify) | (specify) |
| ☐Image contrast | (specify) |
| □Artefacts | (specify) |
| ☐Fat/water homogeneity | (specify) |
| ☐Signalto-noise ratio | (specify) |
| Reconstruction software performance | (specify) |
| ☐Signal-to-noise ratio | (specify) |
| ☐Reconstruction software performance | (specify) |

 DOC1547483 (Rev. 7.0)

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Signature of Sponsor Engineering Representative | Date |
|----------------------------------------------------|------------------------|
| Printed Name of Sponsor Engineering Representative | |
| Sample Document | -Not for Study Use |
| Signature of Chaica! Affirs Project: Minager CUI | rent Sponsofpate vided |
| Printed Name of Clinical Affairs Project Manager | nt version) |
| Signature of Principal Investigator or delegate | Date Received |
| Printed Name of Principal Investigator or delegate | |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



# APPENDIX – EXAMPLE OF VESTIGATION AS INGLEUSED IS POSABLE SWADDLELOG

| Date of check-<br>out | Swaddle<br>Number | Check-out<br>Time | Subject<br>Number | Print name of Study<br>Staff checking out<br>swaddle | Study Staff Signature | Date of<br>disposal of<br>swaddle |
|---|---|---|---|---|---|---|
| Example: | | | | | | |
| 17/Jun/2013 | 000 | 08:42 PM | 000 | Jane Smith | | 17/Jun/13 |
| S | amp | le Doci | ume | nt-Not fo | r Study Us | e |
| | (Pla | 95E 115E | e <i>CIII</i> | rei\$nonsi | orprovideo | / |
| | <u> </u> | <u> </u> | | antivaraia | <u> </u> | |
| | | <i>QC</i> | <i>ICUIII</i> | entversio. | <del>9)</del> | |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



## APPENDIXO - EXAMPLE OF POSSIBLOFTWARE COMPONENTS

The software components listed below are an example of what may be used in subject scanning under an approved MR Procedure Docume per the device configuration management and study protocol.

| 3-Plane Pulse Sequence Family | Spectroscopy PSD Family |
|---|---|
| FGRE | PROBEPRESS CSI single voxel |
| FIESTA | PROBE SVQ (PRESS and STEAM) |
| SSFSE | Gradient Recalled Echo (GRE) Pulse Sequence |
| | Family |
| SEPulse Sequence Family | 2D FIESTA |
| Spin Echo | 2D Fat SAT FIESTA |
| IR | 3D FIESTA |
| Echo Planar Imaging (EPI) Pulsequence Family | 3D FIESTA with fat SAT |
| DW EPI including Focus | 3D FIESTAC |
| DW EPI Tensor | Fast GRE/SPGR (2D and 3D) |
| GRE EPI | 2D GRE/SPGR (2D and 3D) |
| SE EPI | FGRE Time Course |
| One-click applications | 2D FGRE with IR Pr@DMDE) |
| 3DASL | LAVA |
| BRAVO | 2D MERGE |
| CineIR | SWAN |
| Silenz | ASSET Calibration |
| | Fast B1map |
| Fast Spin Echo Pulse Sequendemily | Vascular Pulse Sequence Family |
| FRFSEXL | 2D Fast Phase Contrast |
| FSE IR | 2D Phase Contrast with Cine Mode |
| FSEXL | 3D Phase Contrast |
| FSEXL Double/Triple IR | 2D TOFGRE/SPGR |
| SSFSE | 2D Fast TOFGRE/SPGR |
| | 3D TOFGRE/SPGR |
| T1 FLAIR | 3D Fast TOÆRE/SPGR |
| T2 FLAIR | fAstCINE |
| 3D Cube | FastCINE PC |
| 3D Cube FLAIR | Inhance 3D Velocity |
| 3D FSE | |
| 3D FRFSEXL | |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Visualization | Imaging Options |
|-------------------------|---------------------------|
| FuncTool DTI/FiberTrak | ARC |
| FuncTool DWI/eDWI | ART |
| FuncTool3DASL | ASSET |
| FuncTool Fusion | Blood Suppression |
| FuncTool Spectro | Bright Blood (ASL) |
| Func Tool SER | Cardiac Gating/Triggering |
| FuncTool MR Standard | Classic |
| Volume Viewer: IVI | DE Prepared |
| Volume Viewer: Reformat | Extended Dynamic Range |
| Volume Viewer: 3D View | Flow Compensation |
| SAGE | Fluoro Trigger |
| SR Viewer | fMRI |
| Functool FMRI | IR Prepared |
| Viewer | Mag Transfer |
| Clariview | Multi-Phase |
| Add-Sub | No Phase Wrap |
| Flow Analysis | Phase Sensitive |
| Pasting | RealTime |
| | Sequential |
| | Tailored RF |
| | ZIP 512 |
| | ZIP 1024 |
| - | ZIP x2 |
| | ZIP x 4 |
| | Grad Warp |

Study Number: 114-2014-GES-0035

Protocol: 7.0



## APPENDIX EEXAMPLE OFFIR SCAN LOG

The MR scan log will detail all scanning in this study and from other approved studies that use the same investigational MR device. Enter not applicable ('N/A') for fields that do not apply.

| | ame investigational MR device. Enter not applicable ('N/A'') for fields that do not apply. | | | | | |
|---|---|---|---|---|---|---|
| Scanner<br>Generated<br>Exam<br>Number | Date of<br>Scanning<br>(DD/Mmm/YYYY) | GES/IIR<br>study<br>number<br>(N/S for<br>service,<br>training,<br>etc.) | Subject<br>Number | MR Procedure Document Version (GES only, N/A for IIR/ service, training, etc.) | Anatomy<br>Imaged<br>(N/A for<br>phantoms) | Comments |
| | Samp | e Doo | ument- | <ul><li>Not for</li></ul> | Study l | Jse |
| | (Please | mosti | ise_cur | rentSpon | SOFPIOL | <u>vided</u> |
| | , | <del></del> | <del>scumer</del> | nt-versior | ) | |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



# APPENDIX FEXAMPLB.0TNEONATALMRI INVESTIGATIONAL DECEUSER EXPERIENCE QUESTICANRE

This survey will be completed by an experienced scan operator once for earth Procedure Document Phase 1 and once at the end of Phase 2.

These survey questionwill be completed by the scan operator for each patient on a scale of to 5 or marked as 'not applicable' (N/A) follows:

- 1 = strongly disagree
- 2 = disagree
- 3 = neither agreenor disagree
- 4 = agree
- 5 = strongly agree

Regarding your overall experience with the 0TNeonatal MR investigational device, please rate each of the following on al-5 scale

- 1. I think that I would like to use this system frequently
- 2. I found the system unnecessarily complex
- 3. I thought the system was easy to use
- 4. I think that I would need the support of a technical person to be able to use this system
- 5. I found the various functions in this system were well integrated
- 6. I thought there was too much inconsistency in this system
- 7. I would imagine that most people would learn tose this system very quickly
- 8. I found the system very cumbersome to use
- 9. I felt very confident using the system
- 10. I needed to learn a louf things before I could get going with this system
- 11. I feel confident this system will meet my patient's needs
- 12. How likely is it that you would recommend this product to other professionals in your field?

Sample Document-Not for Study Use

(Please usenost current Sponsorprovided document version)

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



This survey will be completed by an experienced scan operator once for eMM Procedure Document n Phase 1 and once at the end of PhaseResponses should consider the user's overall experience with the 3.0T Neonatal MRthvestigational device.

#### **Questionnaire Instructions**

Please take your time and carefully indicate your responses in the following scales below. PAY ATTENTION TO THE FACT THAT THE SCALES CHANGE their anchor points drittlet left columns from one question to the next. This is done in an effort to reduce bias in the results.

Based on your experiences interacting with the product how would you describe the product?

| | | 4 | 0, | _ | ٠, | ٥, | 4 | |
|-----|-------------|---|----|---|-----|-----|-------|---------------|
| 1) | Learnable | O | O | 0 | · O | · O | - O O | Not Learnable |
| 2) | Inefficient | O | 0 | 0 | · O | · O | - O O | Efficient |
| 3) | Resistant | O | 0 | O | -0 | · O | - O O | Responsive |
| 4) | Annoying | O | O | O | · O | · O | - O O | Pleasing |
| 5) | Satisfying | O | O | O | · O | · O | - O O | Dissatisfying |
| 6) | Ineffective | O | O | O | 0 | · O | - O O | Effective |
| 7) | Fast | O | O | O | · O | · O | - O O | Slow |
| 8) | Unfamiliar | O | O | O | 0 | · O | - O O | Familiar |
| 9) | Routine | O | O | O | · O | · O | - O O | Unusual |
| 10) | Easy | O | 0 | O | 0 | · O | - O O | Difficult |
| 11) | Useful | O | O | O | · O | · O | - O O | Useless |
| 12) | Bad | O | O | 0 | · O | O | - O O | Good |

Sample Document-Not for Study Use

(Please usenost current Sponsorprovided document version)

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



# APPENDIXG-EXAMPLE OSINGLEUSE DISPOSABISWADDLEUSER EXPERIENCE QUESTIONIRE

These assessments are designed to assess the usability the single-use disposable swaddle component associated with the 3.0T Neonatal MRI investigational device on a per patient basis. This survey will be completed by the scan operator for each patient that uses a swaddle.

These survey questions will be completed by the scan operator for each patient on a scale of 1 to 5 or marked as 'not applicable' (N/A), as follows:

- 1 = strongly disagree
- 2 = disagree
- 3 = neither agree nor disagree
- 4 = a gree
- 5 = strongly agree

Regarding your overall experience with the Single-use Disposable Swaddle device, please rate each of the following on a 1-5 scale:

- 1. I think that I would like to use this swaddle frequently
- 2. I found the swaddle unnecessarily complex
- 3. Ithought the swaddle was easy to use
- 4. Ithink that I would need the support of a technical person to be able to use this swaddle
- 5. I found the various functions in this swaddle were well integrated
- 6. Ithought there was too much inconsistency in this swaddle
- 7. I would imagine that most people would learn to use this swaddle very quickly
- 8. I found the swaddle very cumbersome to use
- 9. I felt very confident using the swaddle
- 10. Ineeded to learn a lot of things before I could get going with the swaddle
- 11. I feel confident the swaddle will meet my patient's needs
- 12. How likely is it that you would recommend the swaddle to other professionals in your field?

Sample Document-Not for Study Use

(Please us**e**nost current Sponsorprovided document version)

Study Number: 114-2014-GES-0035

Protocol: 7.0



#### **Questionnaire Instructions**

Please take your time and carefully indicate your responses in the following scales below. PAY ATTENTION TO THE FACT THAT THE SCALES CHANGE their anchor points in the left and right columns from one question to the next. This is done in an effort to reduce bias in the results.

Based on your experiences interacting with the product how would you describe the product?

Somewhat
Sightly
Sightly
Somewhat
Extremely

| 1) Routine | OO | OO- | O | OO | Unusual |
|----------------|---------|-------|--------|----------|---------------|
| 2) Inefficient | OO | OO- | O | OO | Efficient |
| 3) Irrelevant | OO | OO- | O | OO | Relevant |
| 4) Annoying | OO | OO- | O | OO | Pleasing |
| 5) Satisfying | OO | OO- | O | OO | Dissatisfying |
| 6) Ineffective | OO | OO- | O | OO | Effective |
| 7) Fast | OO | OO- | O | OO | Slow |
| 8) Unfamiliar | OO | OO- | O | OO | Familiar |
| 9) Learnable | OO | OO- | O | OO | Not Learnable |
| 10)Easy | OO | OO- | O | OO | Difficult |
| 11)Useful | OO | OO- | O | OO | Useless |
| 12)Bad | OO | OO- | O | OO | Good |
| Sa | mple Do | cumer | nt-Not | for Stud | ly Use |


Study Number: 114-2014-GES-0035

Protocol: 7.0



## APPENDIX H: AMENDMENTO PROTOCOL VERISIOO

**Purpose** This amendment document describes the changes from protocol version 1.0 to 2.0 to account for change in Sponsor medical monitor.

The following amendments were made to version 1.0 to produce version 2.0. Point-by-point revisions are shown as additions in double-underline (double-underline) and deletions in strikethrough (strikethrough) for each change made in this amendment for the previous version.

| Item | Section | Revision or Clarification | | Justification |
|---|---|---|---|---|
| 1 | Study synopsis | Medical Monitor Name:-<br>Reee Lazebnik<br>Jeff Hersh MD | Address: 3200 N Grandview Blvd Waukesha, WI 531881678 Telephone:+1-262-366- 7295262-312-1407 E-mail: Roee.Lazebnik@ge.com Jeff.Hersh@ge.com | Updated amendment<br>version to reflect<br>change in Sponsor<br>medical monitor. |
| 2 | Section 10.4. Management of Serious Adverse Event and Unanticipated Adverse Device Effect Reporting | <del>Roce</del><br>+1- <del>262</del><br>/ | ntact for SAEsand/or UADEs Lazebnikleff Hersh MD 422 5126262-366-7295 Fax 800-888-3983 Fmail: SAE@ge.com | Updated amendment version to reflect change in Sponsor medical monitor. |

Study Number: 114-2014-GES-0035

Protocol: 7.0



### APPENDIX I: AMENDMENTO PROTOCOL VERSI200

Purpose This amendment document describes the changes from protocol version 2.0 to 3.0, as follows:

- 1. To clarify that the primary endpoint of the study is in accordance with Section 2.1 of Annex Xof the EU Medical Devices Directive, which species that verification of performance across the study cohort is an essential requirement of the study.
- 2. To clarify that the planned duration of the study is 24-months, in accordance with requirements of ISO14155.
- 3. To add the feed and sleep procedure, as required by the local site IRB in accordance with the site standard of care requirements.

The following amendments were made to version 2.0 to produce version 3.0. Point-by-point revisions are shown as additions in double-underline (<u>double-underline</u>) and deletions in strikethrough (strikethrough) for each change made in this amendment for the previous version.

| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 3 | STUDY SYNOPSIS | This is a twephase prospective clinical studgevaluating the performance and safety of the investigational MRI device for neonates and infants including: Images, associated image data, and subject data collected in bo phases of this study may be used for future engineering development and activities that support MR product developmen including Sponsorauthorized scientific and marketing activities. Images and associated data from Phase 2 are intended for use a samples fo@ummary evaluation of safety and performance from Phase 1 and Phase 2 may be used in supportrefgulatory submission including filings for European CE marke cehert based analyses are planned for any phase of this study Duration: The study plans to actively enrol patients for approximately 24 months. | that the primary objective of the study is analysis of performance and safety of the device. In accordance with ISO14155, the 24 month planned duration of the study |
| 4 | Section 2.1.2. 3.0T<br>Neonatal MRI<br>Investigational Device<br>Components and Initial<br>Configuration | System Service Toolehantoms (Simulations): | is specified. Corrected typographical error of omitted punctuation ("/" mark). |
| 5 | Section 3.1. Hypothesis | There is no statistical hypothesis being tested in this study. <u>Descriptive statistics will be used to provide summary evaluation of performance and safety data</u> . | Clarified that an evaluation summary using descriptive statistics is required for EU regulatory submission. |
| 6 | Section 3.2. Justification | This study is beig done in two parts to optimize and collect data from a new MRI device for use in neonates and infants, the 3.0T Neonatal MRI investigational device. The first part of this study is being conducted to demonstrate the feasibility of attaining diagnostic quality images and data using the 3.0T Neonatal MRI | Clarified that an evaluation summary using descriptive statistics is required |

**Study Number:** 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | investigational device in neonates and infants with various hardware and software configurations. The second part of this study is being conducted to collect images and associated data i neonates and infants from a fixed hardware and software configuration of the 3.0T Neonatal MRI investigational device in support of regulatory activities in the European Union (EU), including CE markSummary performance and safety evaluations from both parts of the study may be disclosed to regulatory agencies as part of this study. | for EU regulatory submission. |
| 7 | Section 3.3.1. Primary<br>Objective(s): | Toevaluate the safety and performance of the device by collection of collectimages and associated data using the 3.0T Neonatal M investigational device that demonstrates the feasibility of use in clinical neonate and infant populations. | Per MHRA requirements in Annex 1 Section 2.1 of EU Medical Device Directive, clarified that the primary objective of the study is analysis of performance and safety of the device. |
| 8 | Section 3.4.1. Primary endpoints | For both Phase 1 and Phase 2, primary endpoints will be orded as: Collection of MR images and associated data per quotas (Section 5.1.1 - Quotas by Anatomic Region) Performance will be determined by proportion of images determined to be of evaluable or non-evaluable diagnostic quality Safety will be determine by summary rates of adverse events | Clarified the primary endpoint performance and safety measures, in accordance with revised objective described above. |
| 9 | Section 3.4.2. Secondary endpoints | MR image quality evaluation(s), per-phase as follows: Phase 1 and 2 (all subjects): Overall image quality rated on a 15 Likert scale Phase 1 Qualitative evaluation and optimization (Summary Report) provided by PI, asper applicable MR Procedure Document Phase 2-Evaluations as described in the MR Procedure Document | Clarified that engineering performance endpoints are secondary. Per EU Annex X requirements, a measure of overall quality is required for all subjects in the study. The appendix is revised to clarify that this measure is required for all subjects in Phase 1 and Phase 2. |
| 10 | Section 4.1.1. Study Typ | This is a twophase, singlesite, openlabel, prospective research study involving human neonate and infant subjects. Here will be no comparative or cohortbased statistical analyses of efficacy or safety, and therefore no randomization. This study is designed as two-phase clinical trial with an adaptive feasibility and | Clarified that an evaluation summary using descriptive statistics is required |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | optimization phase (Phase 1) and controlled image collection stu (Phase 2). Phase 1 is being conducted to optimize and calibrate the device subsequent data collection in Phase 2 of this studyBoth parts; which is being done formay be used for regulatory submission purposes, including CE mark and submissions to other global regulatory authorities in other countries. Not Randomization is not required, as randomi there are is no comparative analyses typothesis testing | for EU regulatory<br>submission. |
| 11 | Section 4.1.2. Rationale<br>for Two-Phase Study<br>Design | Phase 2 Phase 1 will be followed by a sequential second phase (Phase 2) to collect human images and data intended to as sami images and associated pesubject data for use in regulatory submissions. No comparative or cohort based analyses will be conducted on this population as part of this study. | Clarified that an evaluation summary using descriptive statistics is required for EU regulatory submission. |
| 12 | Section 5.8 Duration of<br>Enrolment | 5.8 Duration of Enrolment The study plans to actively enrol patients for approximately 24 months. | In accordance with ISO14155, the 24 month planned duration of the study is specified. |
| 13 | | Phase2 will be conducted to collect sample images and associated data for regulatory submission No cohort based analysis is intended for this population, and data will only be recorded and stored on a pesubject basis. While hardware and software may be modified throughout Phase 1, a fixed hardware and software configuration will be used for all Phase 2 scanning. Based on the results of Phase MR Procedure Document (si) be provided to the site and used consistenting all Phase 2 scanning. | Clarified that an evaluation summary using descriptive statistics is required for EU regulatory submission. |
| 14 | Section 6.3.1. PreMR<br>Scanning Activities | Pre-Study Feed and Sleep Procedures Per the applicable standard of care procedures required at the investigational site, each participating neonate or infant subject will be allowed adequate feed and sleep to ensure minimum disruption of care during MRI scanning, as follows: c. The subject will be either breast or bottle fed by or in the presence of the parent/legal guardian. d. The subject will be placed in a position that is relaxed and comfortable, with the expectation that it will be reasonably possible for the subject to sleep through the MRI scan. | Added site IRB-required feed and sleep procedure, in accordance with local site standard of care requirements. |
| 15 | Section 6.3.4.<br>Evaluations | Image Assessments Evaluations Image Performance Evaluation Image sets will be labeled according to subject identification number. Images will be evaluated as shown in Figure 2. | Added figure to clarify<br>that evaluable/non-<br>evaluable constitutes<br>the primary<br>performance<br>measure. Added<br>clarification that a<br>third reader will |
**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | | arbitrate to produce |
| | | Eligible participant consents and undergoes Neonatal MMI scan Was an image dataset rated evaluable by Pl Assessments (one reader) and co-investigator? Assessments (one reader) | final evaluable/non- |
| | | | evaluable decision for |
| | | No Non-evaluable | inclusion in analyses, |
| | | NO DATA Document reason on CRF Record reason as acquisition | in the event of |
| | | (i.e. withdrawal, technical issue, scheduling, etc.) ssue or image quality issue | disagreement |
| | | | between the Pland |
| | | NON-DIAGNOSTIC DUE TO IMAGE QUALITY NON-DIAGNOSTIC DUE TO IMAGE QUALITY | neonatologist. This is |
| | | ISSUE ISSUE ISSUE (reasons such as withdrawl, technical issue, scheduling, etc. prevented acquisition of some for diagnostic use) | required due to the |
| | | or all target views necessary for diagnostic use) | _ |
| | | Figure 2. Flavorhant of nonforman and available in Detarmination of | addition of summary |
| | | Figure 2—Flowchart of performance evaluation. Determination of used as the primary performance measure. All secondary Image Q | |
| | | | 1 |
| | | MR image datasets for each subject will be evaluated twice, once | submission for CE |
| | | by the Principal Investigator and once by the neonatologist co-<br>investigator or authorized designee as: | mark of the device in |
| | | | accordance with the |
| | | Evaluable (Diagnostic Quality), or | EU Medical Device |
| | | Non-evaluable (Non-Diagnostic quality). | Directive. |
| | | The printed name and signature of the image evaluator(s) will be | |
| | | recorded. In the event that the two readers disagree on whether | |
| | | an image is evaluable or non-evaluable, a third medically qualified | |
| | | reader will arbitrate to provide an evaluable/non-evaluable decision, which will be recorded to the CRF and treated as the final | |
| | | decision for the image set. | |
| | Section 8.1.2. Statistical | | |
| 6 | | Images and associated data being collected in this study are | Clarified that an |
| | Analysis Methods | intended for use on a per-subject basis. Asummary evaluation of | evaluation summary |
| | | primary performance and safety endpoints and, if necessary, secondary image quality assessments will be prepared by the | using descriptive |
| | | Sponsor and includes in the final clinical study report. Descriptive | statistics is required |
| | | statistics may, as necessary, be used to summarize relevant | for EU regulatory |
| | | results. This evaluation may be used for regulatory submission | submission. |
| | | purposes. | |
| | | No cohort-based analyses or descriptive summaries will be | |
| | | provided for any endpoint as part of this study. Upon completion of | |
| | | this study, the Sponsor's authorized research and engineering | |
| | | program may utilize data collected in this study in full or in part for | |
| | | authorized engineering purposes. | |
| 17 | Section 9.0 OTHER | 8.5.9.0 OTHER INTERIM ACTIVITIES (QUALITATIVE INTERIM | Assigned separate |
| | INTERIM ACTIVITIES | SUMMARIES) | numbering to this |
| | (QUALITATIVE INTERIM | l | section to clearly |
| | SUMMARIES) | 8.5.1.9.1 Phase 1 Qualitative Investigator Summary | indicate that these |
| | / | | additional activities |
| | | 8.5.2.9.2 Phase 1 and Phase 2 Endf-Phase Interim Reports | |
| | | | are not part of |
| | | | statistical analysis |
| | | | (Section 8 and its sub- |
| | | | sections). |
| | | | Correspondingly, |
| | | | attached sub-sections |
| | | | assume headings |
| | | | beginning with 9.X |
| 1 0 | Section 8.3 Handling of | 8.4 8.3 Handling of Missing Data | |
| 18 | Missing Data | O.T. STATE I INITIAL OF IMPOSING DAMA | Clarified that an |
| | IVIISSIII Data | | evaluation summary |

**Study Number:** 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | There are no cohortbased analysed he Sponsor may descriptive summarize the primary performance and safety endpoints from Phase 1 and Phase 2 of this study the Sponsor observed that the dataset for any subject is incomplete, additional clarification from the investigator may be requested. The Sponsor may additionally request copies of any clinical imaging datasets (including MRI so datasets and other clinically indicated imaging examinations) that are conducted as followup to unexpected findings observed in this study. | statistics is required<br>for EU regulatory<br>submission.The<br>section is renumbered |
| 18 | Section 84 Pass/Fail<br>Criteria of the Study | 8.5 8.4. Pass/Fail Criteria of the Study The study will be considered successfuls in the study will be considered successfuls in the study will be considered successfuls in the study will be considered successfuls in the study will be considered successful to the study of the | Clarified that an evaluation summary using descriptive statistics is required for EU regulatory submission. The section is renumbered due to above explained separation of statistical and nonstatistical sections into separate Sections 8 and 9, respectively, for clarity of original protocol intent. |
| 19 | APPENDIX BEXAMPLE OF MR PROCEDURE DOCUMENT | Overall Image Quality (required for all subjects) Other Engineering Performance MeasuresPerformance | Per EU Annex X requirements, a measure of overall quality is required for all subjects in the study. The appendix is revised to clarify that this measure is required for all subjects in Phase 1 and Phase 2. |
| 20 | Throughout | Updated US English spelling conventions to conventional UK Enspelling and MS word style throughout. No atges other than spelling were made throughout as part of this amendment, other than those documented in this appendix. | |
| 21 | Throughout | Removed the "Adaptive" throughout. | Per differences regarding implementation of |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0





| Item | Section | Revision or Clarification | Justification |
|------|---------|---------------------------|------------------------|
| | | | adaptive trialsin the |
| | | | EU, US, and other |
| | | | global regions, the |
| | | | term "adaptive" was |
| | | | determined to be |
| | | | misused in this |
| | | | context and could be |
| | | | misleading that the |
| | | | study is statistically |
| | | | adaptive (rather than |
| | | | adaption of iterative |
| | | | engineering |
| | | | parameters,as per |
| | | | protocol intent). This |
| | | | term is removed |
| | | | throughout to clarify |
| | | | the original protocol |
| | | | intent, and does not |
| | | | reflect a change in |
| | | | study design or risk |
| | | | level. |

Study Number: 114-2014-GES-0035

Protocol: 7.0



## APPENDIX: AMENDMENT TO PROTOL VERSION 3.0

**Purpose** This amendment document describes the changes from protocol version 3.0 to 4.0, as follows:

- 1. To clarify that MR system log files containing operating parameters relevant to device safety and performance models are being routinely collected for all study scanning.
- 2. To update references, symbols, and terminology, as requested for clarification purposes by the MHRA

The following amendments were made to version 3.0 to produce version 4.0. Point-by-point revisions are shown as additions in double-underline (double-underline) and deletions in strikethrough (strikethrough) for each change made in this amendment for the previous version.

| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 22 | Investigator's Signature<br>Page | I hereby agree to: (i) Conduct the investigation in accordance with the agreement, the investigationalplan, applicable MHRA or applicable government regulations, and conditions of approval imposed by the reviewing Ethics Committee, IRB or governing regulate body: (ii) Supervise all testing of the device involving human subjects; and (iii) Ensure that the requirements for obtaining informed consent are met. | Updated required language for investigator signature pages, as per current Sponsor global template requirements. These changes are applicable for all clinical trials conducted by the Sponsor. |
| | | <u>I have read this protocol and study related documents and agree</u><br>to conduct this study in full accordance with the stipulations of the<br>protocol described herein, and any subsequent amendments. | |
| 23 | Synopsis:<br>Device/Product<br>Description | Small-footprint 3.0T NeonataMRI investigational device capable being located in a NICU and its componentincluding a neonate/infant single-use disposableswaddle | Updated language for consistency with the terminology found in the body of the protocol. |
| 24 | Section 1.2. Literature<br>Review | In particular, neonatal MRI has become standard clinical care for neurological and orthopaedic applications at many clinical facilities; <sup>2</sup> <sub>-</sub> <sup>3</sup> <sub>-</sub> <sup>4</sup> <sub>-</sub> <sup>5</sup> | Added citations to support this statement. |
| 25 | Section 1.4.1. Risks | While serious adverse events can occur in MRI exams in rare cases, typically with adverse events occurring as a result of then failure to correctly follow routine site MR safety rocedures for scanning are not correctly followed no serious adverse events are anticipated in this study. | Clarified the language, as per original intent of the statement. |
| 26 | Section 2.1.1. 3.0T<br>Neonatal MRI<br>Investigational Device | This device includes and MR system | Correction to spelling (typographical) |
| 27 | Section 2.1.2. 3.0T<br>Neonatal MRI<br>Investigational Device<br>Components and Initial<br>Configuration:4. | The transmitting and receiving coil is a single channelceive only sixteen rung "birdcage" coil (inner surface accessible to the subject) | Clarified that the coil is for both transmit and receive functions. |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | Radiofrequency (RF)<br>System | | |
| 28 | Section 2.3Risk<br>Category and Rationale | The MRI device used in this study uses static magnetic field strengths <4.0T, which are widely accepted to pose minimal risk to typical adults, children, and infants/neonatepatients as detailed in the US FDA Guidan@riteriafor Significant Risk Investigations of Magnetic Resonance Diagnostic Devares contemporary medical literature comparable with routine clinical MRI examination <sup>26,27</sup> | Clarified and added citation. |
| 29 | Section 2.3.1. MR Safe,<br>Conditional, and Unsafe | Label Description (typical use) MR or MR Safe MR | Updated symbols to<br>current version of<br>ASTM F2503. |
| | | MR Conditional MR Unsafe | |
| | | MR Safe: Devices with scientific rationale or test data indicating that the device poses no known hazards in all MR environments. MR Conditional: Devices with experimental data indicating that the device poses no known bazards in specified MR environments with specified conditions of usage. MR Unsafe: Devices with scientific rationale indicating that the device is known to pose hazards in all MR environments. | |
| 30 | Section 2.5.5. Maintenance and Replacement: (a) | a. Access device(s)-interson or remotely (such as through TVA/Ti or other secure remote connection) for quality control, trouble shooting, training, realtime image optimization to collect system configuration and system log filesor other purposes required for device maintenance, installationor-de-installation, and/or system data collection. | Clarified that remote<br>access is used as par<br>of routine data<br>collection of MR<br>system log files. |
| 31 | Section 3.2. Justification | This study is being done in two parts to optimize and collect data from a new MRI device for use in neonates and infants, the 3.0T Neonatal MRI investigational device. The first part of this study is being conducted to demonstrate the feasibilit <u>and safety</u> of attaining diagnostic quality images and data using the 3.0T Neonatal MRI investigational device in neonates and infants with various hardware and software configurations. The second part of this study is being conducted to collect images and associate data in neonates and infants from a fixed hardware and software | operating parameters contained in system log files, such as SAF data, will be routinely collected as part of this study. |

 DOC1547483 (Rev. 7.0)

Version Date: 25/Sep/2015

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | configuration of the 3.0T Neonatal MRI investigational device in support of regulatory activities in the European Union (EU), including CE markMR system log files containing operating parameters relative to safety and performance calculations will be systematically collected throughout the study for all subjects. Summary performance and safety evaluations from both parts of the study may be disclosed to regulatory agencies as | |
| 32 | Section 3.4.1. Primary endpoints | Safety will be determin <u>d</u> by summary rates of adverse events | Correction to spelling (typographical) |
| 33 | Section 5.3.1. Vulnerabl<br>Subjects | The Sponsor has conducted previous internal testing using phantoms to confirm evaluate the safety of the device for use on humans. | Updated terminology for consistency with internal Sponsor documentation. |
| 34 | Section 6.1.1. Quality<br>Control Scans | The device is equipped with a predictive SAR model designed to conservatively limit actual SAR exposure in research subjects. T predictive SAR model used on the system is detailed in the technical documentation for the Neonatal MRI device. Each scan session will include sequences designed to generate a range of actual SAR data which is stored imay besystem logs and subsequently collected by the Sponsor's engineering representatives from system data and logs of study procedures Throughout the study, system log files containing experimentally generated SAR data will be routinely collected, along with relevance clinical data such as patient weight as described in subsequent protocol sections, necessary for future evaluation of the system's predictive SAR model versus actual clinical data in the infant/neonate population. SAR levels will not exceed levels of 4 W/kg Whole Body, 3 W/kg | system log files containing operating parameter data, including SAR data, will be routinely collected. This data is intended for use in evaluating |
| 35 | Section 6.3.2. MR<br>Scanning Procedures:<br>MR Scanning<br>Information | Anatomy scanned (i.eneurological (head/neck/spine) cardiac/thorax, or abdominal/pelvis) | Corrected erroneous statement. All scanning in this protocol is of the neurological (head/neck/spine) anatomy. Other studies are being concurrently conducted by the Sponsor that examine additional anatomy types. |
| 36 | Section 11.1. Foreseeable Adverse Events and Device Effects | Peripheral Nerve Stimulation: Transient skin sensations ('tingling' or peripheral nerve stimulation (PNS) is relatedd b/dt and gradient rise time, and isexpected to be rare in neonates and infants due to small skin surface area and conservative device thresholds: Subjecting infants to sudden, rapidly changing gradient magnetic fields during imagig can, induce circulating currents in conductive tissues of the body that typically are not | Clarified PNS risk as<br>per current medical<br>literature, including<br>citations. |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | painful and resolveResolution is typically pontaneously though, in theory, discomfort or pair rare cases can cause discomfort pain injury from PNS in infants possible. 26 or death. | |
| 37 | References | 2. Malik S, Beqiri A, Price A, Teixeira J, Hand J, Hajnal J. Specifiabsorptionrate in neonates undergoing magnetic resonance procedures at 1.5 and 3T. NMR Biomed. 2015;28(3):382. 3. Glass H, Bonifacio S, Sullivan J, et al. MRI and Ultrasound Inperterm Infants with Seizures. J Child Neurol. 2009;24(9):41103. 27. Schenck J. Safety of Strong, Static Magnetic Fields. J Mag R. Img. 2000;12:219. 28. Alibadi F, Askary R. Effects of Tadkilbesthetic Stimulation on Low Birth Weight Neonates. Iran J Pediatr. 2013;23(3):299. 29. Anbeek P, Vincken K, Groenendaal Fritane, van Osch M, van der Grond J. Probabilistic brain tissue segmentation in neonatal magnetic resonance imaging. Pediatr Res. 2008;63(2):638 | support the added citations in the document, and renumbered references appropriately in order of sequential appearance in the document. |

Study Number: 114-2014-GES-0035

Protocol: 7.0



## APPENDIX K: AMENDMENTO PROTOCOL VERISIA 0

Purpose This amendment document describes the changes from protocol version 4.0 to 5.0, as follows:

1. To clarify body temperature measurement and associated procedures for setup and calibration of the Invivo Expression monitor for monitoring of body temperature during MRI scanning.

The following amendments were made to version 4.0 to produce version 5.0. Point-by-point revisions are shown as additions in double-underline (<u>double-underline</u>) and deletions in strikethrough (<u>strikethrough</u>) for each change made in this amendment for the previous version.

| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 38 | Section 2.1.4. Other MR<br>Equipment | Invivo Corp patient monitors will be used during study procedures to monitor subject vital signsbody temperature (on the Expression Monitor using a singlese sensor) and O <sub>2</sub> saturation. | Added text to clarify the original intent that body temperature ismeasured during scanning using the MRI compatible Expression Monitor. |
| 39 | Section 6.3.1. PreMR<br>Scanning Activities | Pre-sean Transport Subject Information The following prescan session subject information will be recorded for all subjects: • gender • age since birth (days for subjects aged ≤30 and months for subjects aged >30 days) • gestational age (for subjects ≤30 days old) • infant or neonate status (neonate = birth to ≤30 days; infant >30 days to <2 years) • Pre-transport temperature body temperature measured just before leaving the incubator or crib, measured according to the standard clinical practice at the investigational site stollows: • temperature-measurement value • device type (Expression Monitor [Invivo] or standard of care device), and • anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify) | device type, and anatomical area for temperature measures in the pretransport period. |
| 40 | Section 6.3.1. Pre-MR<br>Scanning Activities | Preparation for Scanning Immediately before initiating the scan, ensure that the Expression Monitor (Invivo) is connected and monitoring vital signs, including but not limited to body temperature and O2 saturation. Once acclimated to the scan environment, the following scanning information shall be recorded by the scan operator, including the following: • Prescanning baseline temperature ody temperature measurement made with an Expression Monitor (Invivo), as follows: | Added a new temperature measurement during the period in the MRI area immediately before scanning, This is collected as a baseline for confirmation that the subject's body temperature does not exceed 0.5°C during scanning. All temperature measures during scanning |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0





| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | <ul> <li>the time (minutes) allowed for acclimation once in the magnet bore before taking the temperature measurement</li> <li>temperature measurement value</li> <li>anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify)</li> <li>The study staff will set the alarm level on the Expression Monitor (Invivo) to trigger at 0.5°C above the pre-scanning baseline temperature.</li> </ul> | will be taken using the Invivo<br>Expression Monitor that is<br>MRI compatible. |
| 41 | Section 6.3.2. MR<br>Scanning Procedures | Monitoring Subjects During MRI Scanning During MRI scanning, subjects will be monitored in real-time using a properly functioning Expression MRI Patient Monitor (Invivo, Corp; Orlando, FL, USA). The subject will be observed all times during the MR scan by a qualified medical professional (nurse, neonatologist, and/or other medical doctor qualified for neonatal/infant care) on the study staff who shall remain in the magnet room with the subject during scanning. The observing staff should remain in a position where they can readily observe the subject and monitor and, if necessary, contact the scan operator during the scanning session. Aconservative threshold for body temperature alarm is selected, as such that body temperature change is sufficient to trigger an alarm (0.5°C above the pre-scanning baseline temperature) is not in itself considered a clinically significant risk to patients; these patients will be evaluated by a medically qualified member of the study staff for any other possible signs or symptoms and they will determine whether an AE has occurred as per the standard procedures described in Section 11 — Complaint Handling and Adverse Event Reporting. If a body temperature alarm on the monitor is triggered at any time during scanning, the study staff should stop the scan series. Then, the following elements will be documented as part of study data for each such alarm occurrence: • the time of alarm • Alarm Temperaturethe body temperature at time of alarm, based orbody temperature measurement made withan Expression Monitor (Invivo) as follows: • temperature measurement value • anatomical area of measure (specific area of skin surface, i.e., axillary or specify; oesophageal; or other, specify) • the time it takes to return to pre-scanning baseline temperature (minutes/seconds) | Describes that scanning will end if the temperature alarm indicates that body temperature rose more than 0.5°C during MRI scanning, and documents applicable temperatures and if the scan was able to be successfully continued upon resolution of temperature rise. Added that the actual body temperature at alarm and, if applicable, upon continuing the scan will be captured. It is clarified that the 60 minute scanning window only refers to the scanning time in the MR device, and not to setup or preparation time, |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0





| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | Note. In the event that the baby's body temperature does not return to a level at or below the pre-scanning baseline temperature within the study scanning period (not to exceed 60 minutes from first localizer to end of scanning), the patien will be discontinued from the study. | |
| | | o any conditions observed that possibly contributed to temperature rise, such as swaddling, environmental conditions, distress, or scanning conditions? (WN, if yes explain) o decision to continue the scan session (do not continue after first alarm)? (WN) Continuing Temperaturæhe body temperature at the time of scanning wascontinued using an Invivo Expression Monitor, as follows: • temperature measurement value • anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify). Amedically qualified investigator should evaluate each patient to determine if it is safe to continue scanning once the patient's body temperature returns to prescanning baseline temperature or lower in the event of | |
| | | an alarm. If an alarm is triggered more than once during a single scan session, the patient will be discontinued. Subject MR Scanning Procedures The total time that the subject may be in the MR scanner, starting from the start of the first localizer to the time at the end of the last scan; will not exceed sixty (60) minutes. Additional time may be required for setup and removal of the patient. | |
| 42 | Section 6.3.3. Post-scanning MR Procedures | Post-scanning Subject Information Post-scanning information will be recorded for all subjects: • Post-scanning temperatureBody temperature, immediately before removal from the MR scanner (post-scan body temperature) body temperature measurement made with an Invivo Expression Monitor and anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify). • Time of removal from MR device (on 24 hour clock) • Final temperatureBody temperature (measured after transport and just before the subject is moved-placed back into theirthe routine care environment meubator/crib by the same method used for previous body temperature recordings as follows: • temperature measurement value | Differentiated between post-<br>scanning and final<br>temperature measurements. Added specific requirements<br>for capturing the value,<br>device type, and anatomical<br>area for temperature<br>measures in the post-<br>transport period. |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 43 | Section 8.3. Handling of<br>Missing Data | o device type (Expression Monitor [Invivo] or standard of care device), and anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify) Note. It is preferred that the same method as used for the Pretransport Temperature The Sponsor may descriptively summarize the primary performance and safety endpoints from Phase 1 and Phase 2 of this study including the descriptive statistical summar of patients that exhibit a body temperature rise of more than 0.5°C from acclimated prescanning baseline body temperature (resulting in an Expression Monitor alarm during scanning) | Describes intent to include the body temperature in descriptive statistic summary. |
| 44 | Signature Page | | Updated to per current<br>Sponsor procedural<br>requirements. |

Study Number: 114-2014-GES-0035

Protocol: 7.0



## APPENDIX L: AMENDMENTO PROTOCOL VERISIOO

**Purpose** This amendment document describes the changes from protocol version 5.0 to 6.0, as follows:

- 1. To clarify temperature measurement procedures, including that only the MR Safe Invivo Expression monitor may be used during MR scanning and in the MR scan room; standard of care methods may be used for temperature determinations in the patient's clinical care area.
- 2. Clarified that In Vivo Essential monitor is not a required patient transport monitoring system and that site will use their standard of care monitoring system during patient transport. All mention of In Vivo Essential monitor is removed from the protocol.
- 3. To clarify that if scanning is stopped due to alarm, the scanning will be discontinued, but patients may continue on in other parts of the study (i.e. transport) and that data from such subjects may still be used and disclosed to the Sponsor.

The following amendments were made to version 5.0 to produce version 6.0. Point-by-point revisions are shown as additions in double-underline (<u>double-underline</u>) and deletions in strikethrough (<u>strikethrough</u>) for each change made in this amendment for the previous version.

| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 45 | Section 2.1.4. Other MR<br>Equipment | Invivo Corp patient monitor will be used during study procedures to monitor subject vital signsbody temperature (on the Expressio Monitor using a singleuse senso <u>rin the MRI scan roor</u> ); and Q saturation. | |
| | | Essential Monitor (Invivo Corp)This is a patient transport monitoring system. This is MR Conditional patient monitor system labelled for use in neonate and infant populations that may remain the magnet room during scanning if conditions are met. This is a small monitor that attaches to the patient table for transport | |
| | | <del>purposes</del> . | system as per their standard of care. |
| 46 | Section 6.3.1. PreMR<br>Scanning Activities | General Method for Recording Temperature Subject body temperature will be recorded at defined intervals before, during, and after scanning as detailed in the following sections. In the MR suite and during scanning, MR Safe Invivo Expression monitor should be used to determine temperature an other vital signs. | Clarification to when monitor may be used for study temperature measurements. |
| 47 | Section 6.3.1. PreMR<br>Scanning Activities<br>Pre-Transport Subject<br>Information | Pretransport temperature body temperature just before leaving the incubator orcrib, measured according to the standard clinical practice at the investigational site, as follows: temperature measurement value device type (Expression monitor [Invivo] or record standard of care device), and anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify) | Expression monitor is used during MR scanning. Corrected that standard of care temperature measurements will be |
| 48 | Section 6.3.1. Pre-MR<br>Scanning Activities -<br>Pre-scan Environmental<br>Condition | Immediately prior to the first scan series, the following environmental conditions in the MR scanning room will be recorded: Scan room temperature System temperature, per MR device console | Clarified that the<br>system console does<br>not display this<br>temperature and thus<br>it cannot be recorded. |

**Study Number:** 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 49 | Section 6.3.1. PreMR<br>Scanning Activities<br>Preparation for<br>Scanning | Pre-transport temperature body temperature just before leaving theincubator or crib, measured according to the standard clinical practice at the investigational site, as follows: temperature measurement value device type (Expression monitor [Invivo] or record standard of care device), and anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify) | will not perform oesophageal measurements. Corrected that standard of care temperature |
| 50 | Section 6.3.1. Pre-MR Scanning Activities – Duration of Active Enrolment | Active enrolment will be considered to end on a persubject basis upon the later of: a. The time that the subject is returned to his or her standard of care clinical environment-and all Sponsor provided devices are removed from the subject, including Sponsor-provided swaddle, protective padding, and all other study devices OR b. The time that all Sponsor provided devices are removed from the subject, including Sponsor-provided swaddle, protective padding, and all other study devices. b. After active enrolment ends, images and data about any standard of care follow-up or other medical care resulting from unexpected findings may still be accessed observationally and collected by the Sponsor for research purposes. | Clarified end of subject active enrolment in the |
| 51 | Section 6.3.1. Pre-MR Scanning Activities – General Method for Recording Temperature | Subject body temperature will be recorded at defined intervals before, during, and after scanning as detailed in the following sections. In the MR suite and during scanning, MR Safe Invivo Expression monitors should be used to determine temperature and other vital signs. Outside of the MR suite, Invivo Essential monitors should be used to determine temperature and other vital signs. In the event that these monitors are not able to be used for any reason, study temperature measurements may be taken using alternative standard of care body temperature measurement methods, and the type of body temperature measurement method should be documents on the CRF. Temperature and vital signs measurement devices used during scanning or in the MR suite must be labeled as MR Safe or meet the conditions of MR Conditional labelling. | Clarified and simplified the instruction of temperature collection. Clarified that in the MR suite, if for some reason In Vivo Expression monitor is not working, the subject cannot be scanned at all.Outside of the MR suite, other devices can be used to monitor/measure the subject temperature. |
| 52 | Section 6.3.2. MR<br>Scanning Procedures -<br>Monitoring Subjects<br>during MR Scanning | Prescanning baseline temperature ody temperature measurement made with Invivo Expression Monitor (Invivo), as follows: the time (minutes) allowed for acclimation once in the magnet bore before taking the temperature measurement temperature measurement value anatomical area of measure (specific area of skin surface, i.e. a xillary or specify; oesophageal; or other, specify) | Clarified that the site will not perform oesophageal measurements. Also clarified that scanning is discontinued in the event of a larm (subject is not |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0





| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | If a body temperature alarm on the monitor is triggered at any time during scanning, the study staff should stop the scan series Then, the following elements will be documented as part of study data for each such alarm occurrence: the time of alarm Alarm Temperaturethe body temperature at time of alarm, based orbody temperature measurement made with the Expression Monitor (Invivo), as follows: temperature measurement value anatomical area of measure(specific area of skin surfacei.e. axillary or specify; oesophageal; or other, specify). the time it takes to return to prescanning baseline temperature (minutes/seconds) Mota In the event that the baby's body temperature doe not return to a level at or below the prescanning baseline temperature within the study scanning period (not to exceed 60 minutes from first localizer to end of scanning), the patient will be scanning will be discontinued from the study (if collected, the patient's data collected up until this time may still be used for study purposes, and postscanning information may still be recorded about the patient() any conditions observed that possibly contributeto temperature rise, such aswaddling, environmental conditions, distress, or scanning conditions(Y/N), if yes explain) decision to continue the scan session (do not continue after first alarm)? (Y/N) Continuing Temperaturathe body temperature at the time of scanning was continued using aftxpression Monitor (Invivo), as follows: temperature measurement value anatomical area of measure (specific area of skin surface; i.e. axillary or specify; esophageal; or other; specify) Amedically qualified investigator should evaluate each patient to determine if it is safe to continue scanning once the patient to determine if it is safe to continue scanning once the patient to determine if it is as a continued. If collected, the patient's data collected up until this time may still be used for study purposes, and post-scanning information may still be | Corrected that<br>standard of care<br>temperature<br>measurements will be<br>used (Expression is<br>only used in the MR<br>suite. |
| 53 | Section 6.3.3. Post-<br>scanning MR Procedures<br>- Post-scanning Subject<br>Information | Post-scanning information will be recorded for all subjects: • Post-scanning temperatureBody temperature, immediately before removal from the MR scanner (post-scan body temperature), body temperature measurement made with and Expression Monitor (Invivo) and anatomical area of measure (specific area of skin | Clarified that the site will not perform oesophageal measurements. Clarified that Expression monitor is |

 DOC1 547483 (Rev. 7.0) Version Date: 25/Sep/2015

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | surface, i.e. axillary or specificesophageal; or other, specify). Time of removal from MR device (on 24 hour clock) Final temperature Body temperature measured after transport and just before the subject is placed into the routine care environment, as follows: temperature measurement value device type (Expression Monitor [Invivo] or record standard of care device), and anatomical area of measure (specific area of skin surface, i.e. axillary or specify; oesophageal; or other, specify) Note. It is preferred that the same method as used for the Pretransport Temperature Find of Enrolment Time: Time when the patient is returned to the clinical care area and all Sponsor-provided device components (i.e., Swaddle, Invivo monitor, pads, etc.) have been removed from the subject. | used during MR scanning, and Essential Monitor is used during transport (temperature measurements during transport are made according to the standard of care). Corrected that standard of care temperature measurements will be used (Expression is only used in the MR suite. Removed Time of removal from MR device (on 24 hour clock) and clarified end of enrolment time definition. |
| 54 | Section 6.3.3. Post-<br>scanning MR Procedures<br>- Post Scan<br>Environmental<br>Conditions | At the end of the last scan series when the scan operator enters the scan room to remove the subject from the MR device, the scan operator will record: Scan room temperature System temperature, per MR device console | Clarified that the<br>system console does<br>not display this<br>temperature and thus<br>it cannot be recorded |
| 55 | Section 6.5 - Withdrawal and Discontinuation Criteria | All subjects must be admitted for care in the NICU or other neonatal or infant care department or unit affiliated with the investigational site at the time of enrolment and scanning to be eligible to participate in this study. If a subject is discharged from clinical care at the investigational site prior to MR scanning, the subject will be withdrawn from the study. The subject's medical care shall take precedence over any imaging or other procedures associated with the study. If it is determined during the exam that the study imaging will in any way negatively impact required clinical care, the subject shall be immediately withdrawn from the study. In the event the subject appears to be in pain or undue discomfort, if potentially destabilizing vital signs are observed by visual inspection or via monitoring equipment, or if the parent(s) or legally authorized representative requests to discontinue study procedures, the study procedures will be discontinued immediately and the subject will be removed from study—as determined necessary by the medically qualified staffas soon as possible according to the standard of care at the investigational site. The subject shall be removed from the MR environment as soon as safely possible, and, if necessary, care will be provided to the subject to alleviate any discomfort according to the site's standard of care. Data collected up until the time of withdrawal may still be used and disclosed to the Sponsor for research purpose | Clarified that data collected up until the time of withdrawal (even if scanning is discontinued) will be recorded. |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | The subject's parent or legal guardian may withdraw him or her from study participation at any time, for any reason without consequence. | |
| | | The study staff may withdraw a subject at any time for any reaso | |
| | | The reasons for withdrawal and discontinuation formy subject shall be recorded. These will be reported to the Sponsor. | |
| 56 | Section 14.3 Subject<br>Pseudonymisation | All subject data that is sbmitted to the Sponsor will be identified by the use of a unique subject number assigned as an identification code to the Subject, without dedentification. The scan operator will enter the identification number in the system to complete pseudonymisation. The assigned subject identification number in the system to complete pseudonymisation. The assigned subject identification numberill consist of a four digit number and be issued in consecutive order starting with 0001_according to the Sponsor's Data Management Plan (DMP). Each participating site will maintain a subject identification log, which is a list of all subjects who are enrolled in the study, along with their address and medical record number in the event that they must be contacted in the future. | Updated to reference<br>this detailed<br>description of<br>numbering located in<br>the DMP, as per<br>standard Sponsor<br>procedure. |

Study Number: 114-2014-GES-0035

Protocol: 7.0



## APPENDIX M: AMENDMENTO PROTOCOL VERISIOO

**Purpose** This amendment document describes the changes from protocol version 6.0 to 7.0, as follows:

- 1. To clarify that the two (2) radiologists will act as image evaluators (rather than the PI and a neonatologist). This is done to minimize bias, as the PI and neonatologist may be directly involved in study acquisitions based on specific site practices.
- 2. Clarifies the responsibilities of evaluators and readers in this study in figures and flowcharts, for clarity only (this does not change the original intent or design of the study, other than as described in #1 above).
- 3. To clarify the roles of participating physicians and neonatologists in the study procedure and assessments.
- 4. To clarify the procedures for screenings subjects for enrolment and verify MR safety prior to study procedures.

The following amendments were made to version 6.0 to produce version 7.0. Point-by

-point revisions are shown as additions in double-underline (double-underline) and deletions in strikethrough (strikethrough) for each change made in this amendment for the previous version.

| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 57 | Study Synopsis | <b>Duration</b> : The study plans tæctively enrol patients for approximately 24 months. | Removed the descriptor "active" describing the EC/IRE approved protocol as this is not meant to correspond with the "active" enrolment period for AE reporting purposes. This term is removed to clarify this intent. |
| 58 | Section 2.6. Disposition of the Device/Product | When scanning under active EC/IRB approved tudy protocos is empleted, the following actions will be conducted: | Removed the descriptor "active" describing the EC/IRE approved protocol as this is not meant to correspond with the "active" enrolment period for AE reporting purposes. This term is removed to clarify this intent. |
| 60 | Section 4.2.<br>Controls and<br>Minimization of<br>Bias | The following bias control methods are being employed in this study: d. Selection biaswill be limited by consecutively enrolling subjects meeting the inclusion/exclusion criteria e. Spectrum biaswill be limited by using a population expected to be representative of the general population at the investigational site, without regard for gender, race, or ethnicity. f. Reader bias will be limited by ensuring that evaluators and readers making performance assessments are separate radiologists (not the PI or neonatologist). | Described added protections for reader bias by ensuring that the evaluators making image assessments are separate from the principal investigator. |

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 61 | Section 5.4.<br>Inclusion Criteria | Able to safely undergo an MRI scan, as determined the site's coinvestigator neonatologis medically qualified personnet | Clarified that the site would delegate medically qualified personnel, but this wil |
| | | 6. Are of appropriate size and shape to fit into the bore of the magnet, inclusive of all monitoring equipment, if any, necessary forthe subject's routine clinical cares as a standard of care measurement methods, in accordance with site policies | |
| 62 | Section 5.4.<br>Exclusion Criteria | 6. Have parent(s), guardian(s), or legally authorized representative(s) that require that they accompany the subject into the MR environment that have contraindications to the MR environment or would otherwise be put at undue risk or discomfort, as determined by the investigators medically qualified personnel; 8 7. Have any ferrous or electrical items or non-removable medical devices that are not compatible with MR scanning (including devices labelled as MR Unsafe, MR conditional for which the scanning conditions are not met, or without MR safety labelling that does not satisfy site MR safety requirements) that may pose hazards in the MR scanning or MR environment, in the opinion of the Principal Investigator or medically qualified personnel neonatologist co-investigator-in accordance with the site's MR Safety policy; 8. Have any contraindications or could otherwise be expected to experience detrimental effects to safety, well-being, or medical care, as determined by the Principal Investigator or medically qualified personnel neonatologist co-investigator-in accordance with the site's MR Safety policy; 9. Require any scheduled standard of care procedures that are expected to be adversely impacted by participation in this study, in the opinion of the principal investigator; neonatologist co-investigator, or medically qualified delegate personnel; and | Clarified that the site would delegate medically qualified personnel, but this will be done under the supervision of the PI and the Sponsor will not require that this be delegated to the site neonatologist |
| 63 | Section 5.7<br>Screening and<br>Enrolment | 5.7 Screening and Enrolment 5.6.2 Screening for Enrolment Potential subjects will be identified by the Principal Investigator or other qualified site staff. Informed consent will be obtained for those subjects who agree to participate in the study. Subjects will then be screened for enrolment to ensure the subject is eligible to participate per the inclusion/exclusion criteria, as per the judgement of medically qualified personnel. Subjects who do not qualify based on inclusion/exclusion criteria will be considered screen failures. | Clarified screening requirements to specifically indicate that enrolment happens after consent is provided and before any study procedures are performed (including sizing ring). |

<sup>8</sup> If it is not safe for the parent or guardian that wishes to accompany the subject into the MR environment, the parent or guardian may opt not to accompany the subject. In this case, the subject would not be excluded. Subjects would be excluded if it is determined to be potentially unsafe for a parent or guardian to accompany a subject into the MR scan suite, and the parent or guardian is not willing to allow the subject to be scanned alone while he/she waits in another area of the hospital.

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | Once a subject is determined to be eligible per the inclusion/exclusion | |
| | | criteria including providing written informed consent, the subject will be | |
| | | considered enrolled and assigned a subjectumber. Subjects will be | |
| | | screened to ensure that all of the following conditions are met prior to study enrolment: | |
| | | The subject meets the criteria for inclusion/exclusion, including size | |
| | | requirements, | |
| | | Note: At screening, the subject's size will be determinated to the | |
| | | standard of care at the investigational site (e.g. using a tape measure | |
| | | other standard device). After informed consent is attained for the subject, the Sponsoprovided sizing tool will be used to confirm the | |
| | | subject's size as part of <b>M</b> safety screening. | |
| | | Parents(s) or legal guardian(s) provide written informed consent for the subject's participation, | |
| | | The subject and any person(s) accompanying him or her into the MR | |
| | | environment have been successfully screened according to the standal of care MR safety screening procedures at the investigational site(s), | |
| | | , , , , | |
| | | including supplemental screening for patients that are suspected to have metal object on or implanted in their body (i.e. using ha <b>hd</b> ld | |
| | | metal detectors), to ensure that both the subjected any person(s) who | |
| | | wish to accompany the subject into the MR scanning room are eligible | |
| | | for MR scanning. Written documentation will be retained by the site for | |
| | | MR safety screening. | |
| | | If the subject and/or parent or other person that will accompany the subject fail to meet screening criteria, the subject will be considered as | |
| | | subject fail to fried screening chiefla, the subject will be considered as screen failure and will not be considered enrolled. | |
| | | Subjects that meet the screening criteria will be enrolled and will be | |
| | | considered actively enrolled from the time the subject intact will be | |
| | | swaddle, if used, or removed from his or her normal standard of care | |
| | | environment for transport until the subject is returned to his or her star | |
| | | ef care situation and all MR equipment, such as swaddle or padding, is | |
| | | removed. | |
| | | 5.7.1 MR SafetyScreening | |
| | | Screening will be completed for the subject and any person | |
| | | accompanying him or her into the magnet room prior to allowing | |
| | | entrance into the MR scan room. The scan operator will confirm | |
| | | completion of MR safety screening, per standard clinical ptime at the | |
| | | investigational site. In addition, subjects may be screened for the | |
| | | presence of ferrous metallic objects using a handeld metal detector, | |
| | | under the direction of the principal Investigator or delegate. The subject | |
| | | and anyone accompanying the sbject into the MR scan room, will be | |
| | | provided with mandatory hearing protection, such as earlings or ear | |
| | | <u>plugs combined with ea</u> muffs and/or ear plugs, and other protective devices required by site MR safety policies. | |
| | | Enrolled subjects must be confirmet be of acceptable size for MR | |
| | | scanning in this study using the Sponsprovided sizing tool | |
| | | ("horseshoe" shaped ring) with all required attached medical equipmen | |
| | | presentThis is conducted to verify that the subject and all necessary | |
| | | medical equipment can safely fit into the bore of the MR device with | |
| | | normal airflow and without contacting the bore., at the following | |
| | | intervals:Prior to removal from the normal clinical care environment | |
| | | Immediately prior to MRI scanning (by the scan operator or qualified designee) | |
| | | Note: The sizing tool is a study device that may only be used after | |
| | | written informed consent for participation has been attained. | |


**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| 64 | Section 5.7.<br>Duration of<br>Enrolment | The study plans tæctively enrol patients for approximately 24 months. | Removed the descriptor "active" describing the EC/IRE approved protocol as this is not meant to correspond with the "active" enrolment period for AE reporting purposes. This term is removed to clarify this intent. |
| 65 | Section 6.1.1.<br>Quality Control<br>Scans | | Removed he descriptor "active" describing the EC/IRE approved protocol as this is not meant to correspond with the "active" enrolment period for AE reporting purposes. This term is removed |
| 66 | Section 6.3.1. Pre<br>MR Scanning<br>Activities: MRPre-<br>screeening | safely fit into the study device bore with normal airflow and without | enrolment. |
| 67 | MR Scanning | Duration of Active Enrolment (for AE/SAE reporting purposes) Subjects may be transported to the MR suite before or after removal from their incubator, crib, or other standard of care bedding. Subjects will be considered active enrolled (for AE/SAE reporting purposes) in the study on a persubject basis from the time that the | Removed the descriptor "active" describing the EC/IRE approved protocol as this is not meant to |

 DOC1547483 (Rev. 7.0)

Version Date: 25/Sep/2015

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | Sponsorprovided horseshoeshaped sizing tool is used to measure subject size(the first study procedure of MR Proceeding). It is mandatory that the sizing ring is used for all subjects before other stud procedures to ensure that the subject is of proper size for the MR bore | |
| 68 | Section 6.3.1. Pre<br>MR Scanning<br>Activities:<br>Protective<br>Devices/Procedur<br>es | All subjects require mandatory hearing protection that provides a minimum of 22 dB attenuation prior to MR scanningear plugs or a combination of ear plugs and ear muffs, in accordance with site MR Safety Polices). Use of the horseshoeshaped sizing ring to verify that subjects can safe fit into the bore of the MR device is mandatogand should also be performed before transporting the subject out of their clinical care environment immediately prior to scanning. The scan operator or delegate will ensure that the subject meets the criteria for MR scanning according to that it is prefered in this protocoln addition, the study staff may screen subjects and accompanying person(s) for presence of ferrous metallic objects using a hand-held metal detector, under the direction of the principal Investigator or delegate. If new information shows that the subject doe not meet the site MR Safety Policy requirements, the subject will be withdrawn. | |
| 69 | Section 6.3.4. Evaluations: Performance Evaluation | Performance Evaluation Image sets will be labelled according to subject identification number. Images will be evaluateds evaluable (diagnostic) or noewaluable (non-diagnostic) by two evaluators, and then evaluable images will be read for image quality by a separate reades shown in Figure 2. Original Figure 2 Eligible participant consents and undergoes Neonatal MRI scan NON-DIAGNOSTIC DUE TO ACQUISTION QUALITY ISSUE In withdrawal, technical issue, scheduling, etc. prevented acquisition of some or all target views necessary for diagnostic use) NON-DIAGNOSTIC DUE TO ACQUISTION QUALITY ISSUE Issue or image quality is insufficient for diagnostic use) NON-DIAGNOSTIC DUE TO ACQUISTION QUALITY ISSUE Issue or image quality is insufficient for diagnostic use) Revised Figure 2 Non-DIAGNOSTIC DUE TO IMAGE QUALITY (image quality is insufficient for diagnostic use) Revised Figure 2 | Clarified text and Figure 2 to indicate that the PI will not be the study image evaluator, as an additional bias control. |
| | | Non-Diagnostic Due To Acquisition Quality Issue (reasons such as withdrawa), technical issue, scheduling, etc. presented acquisition of some or all target views necessary for diagnostic use) Figure 2— Flowchart of performance evaluation. Determination of evaluation performance measure. All secondary Image Quality Assessm | |

Study Number: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | | Revision or Clarification | on | | Justification |
|---|---|---|---|---|---|---|
| | | MR image datase delegated radiolo Evaluator 2) once neonatologist coi • Evaluab • Non-eva The evaluations and evaluator(s) will be two readers evaluations and evaluations are two life decision as the final decision | | | | |
| 70 | Section 6.3.4.<br>Evaluations:<br>Image Quality<br>Assessments | 1) that may be the | All evaluable images will be further examined by a single reader (Reader ) that may be the PI or a qualified delegated radiologist for image quality on a 1-5 Likert Scale, 10 as follows: | | | |
| 71 | Section 6.6. Study<br>Flowchart (Table 3) | Additional Sponsor- Requested Assessments MR Images and Data Evaluable (Diagnostic) N on-evaluable (Non- diagnostic) Assessment Image Quality Assessments Overall image quality (based on investigator) § experience | #· | Post-<br>Scan | Reader/ Evaluator Assessme nts X(reader only) (defined in MR Procedure Doc) X (access to) X (reader and evaluator s) X (reader only) X (reader only) | Clarified flowchart language around evaluators and readers. This is a clarification of the original intent, as described above. |

<sup>&</sup>lt;sup>9</sup> An image set may be considered of diagnostic quality if it contains images suitable for diagnosis (not all images views are typically required to be diagnostic based on specific scanning circumstances, so long as applicable views necessary for diagnosis are present)

*Note* For image quality assesment, scores of 3, 4, or 5 will be considered diagnostic quality, and scores of 1 and 2 will be considered non-diagnostic quality.

<sup>&</sup>lt;sup>10</sup> Likert Scale of 45, where:

<sup>1 =</sup> Very Poor

<sup>2 =</sup> Poor

<sup>3 =</sup> Neutral

<sup>4 =</sup> Good

<sup>5 =</sup> Excellent

**Study Number**: 114-2014-GES-0035

Protocol: 7.0



| Item | Section | Revision or Clarification | Justification |
|---|---|---|---|
| | | Image | |
| 72 | Section 11.1. Foreseeable Adverse Events and Device Effects | hearing loss/tinnitus typically related to improper hearing protection ca | plugs or a<br>combination of ear<br>plugs+muffs is<br>required |

End ofDocument